# A prospective, multi-center, randomized, and controlled clinical trial for the evaluation of the safety and efficacy of Filtek<sup>TM</sup> Bulk Fill Posterior Restorative in the direct restoration of Class I and II cavities of posterior teeth

# Statistical Analysis Plan

# V1.1

Statistical Analysis Unit: Medical Statistics Department of National

Cardiovascular Center

**Sponsor:** 3M ESPE Dental Products

**Release Date:** March 3, 2020

# **Confidentiality Statement**

The information contained in this document is proprietary and confidential. Without the written permission of the contact of the Sponsor 3M ESPE Dental Products, it is prohibited to copy, disseminate, or otherwise publish the information.

• round enough after cavity preparation

# **SIGNATURE PAGE**

| Study Title: | A prospective, multi-center, randomized, and controlled clinical trial for the evaluation of the safety and efficacy of Filtek <sup>TM</sup> Bulk Fill Posterior Restorative in the direct restoration of Class I and II cavities of posterior teeth | | | |
|---|---|---|---|---|
| Sponsor: | 3M ESPE Dental Products | | | |
| Study No.: | MDI 0102 | MDI 0102 | | |
| Release Date: | March 3, 2020 | | | |
| Version Number: | V1.1 | | | |
| Sponsor/Agent CRO | Title: | Year | Month | Day |
| Principal Investigator | Title: | Year | Month | Day |
| Author of the Plan (NCCD) | Title: | Year | Month | Day |
| Approver of the Plan (NCCD) | Title: | Year | Month | Day |

# **Table of Contents**

| Cnapter | Page No. |
|---|---|
| SIGNATURE PAGE | |
| ABBREVIATIONS AND DEFINITIONS OF TERMS | |
| 1. Introduction | |
| 2.1 Background data of the disease | |
| 3. Overall design of clinical research | |
| 3.1 Trial objective | |
| 3.2 Selection and justification of methodology | |
| 3.3 Evaluation methodology of efficacy | |
| 3.4. Secondary efficacy measures | |
| 3.5 Evaluation methodology of safety | |
| 4. Investigational device/control product | |
| 4.1. Investigational device | 10 |
| 4.2. Control device | 10 |
| 4.3 Indications of the products | 10 |
| 4.3.1 Indications of the investigational device | 10 |
| 4.3.2 Indications of the control device | |
| 5. Subject selection | 11 |
| 5.1 Inclusion criteria | 11 |
| 5.2 Exclusion criteria | |
| 6. General statistical considerations | |
| 6.1 Determination of the sample size and its justifications | |
| 6.1.1 Statistical design (Test of Hypothesis) | |
| 6.1.2 Total sample size | |
| 6.2 Analysis population | |
| 6.3 Determination rules and flow diagram of analysis population data set | |
| 6.4 Missing values, abnormal values, and outliers | |
| 6.5 Significance level and statistical analysis software | 17 |
| 6.6 Consolidation of centers | |
| 7. Statistical analysis measures and methodology | |
| 7.1 Demographic data and other baseline data | 18 |
| 7.2 Operation information | |
| 7.3 Primary efficacy measures | 18 |
| 7.4. Secondary efficacy measures | 19 |
| 7.5 Safety measures | 20 |
| 7.6 Follow-up data | 20 |
| 7.7 X-ray examination | 20 |
| 7.8 Device defects | 21 |
| 7.9 AEs and SAEs | 21 |
| 7.10 Concomitant medication | 22 |

| 8. GENERATION OF STATISTICAL TABLES, LISTS, AND GRAPHS | 23 |
|---|---|
| Fig. 1 Determination flow diagram of the analysis population data set | 23 |
| Table 1 Determination of the analysis population | 24 |
| Table 2 List of subjects who do not receive any investigational device or are in serious deviation to th | e |
| protocol | 25 |
| Table 3 Statistical analysis results of subjects in serious deviation to the protocol (CRF collection | n) 26 |
| Table 4 List of subjects in serious deviation to the protocol (CRF collection) | 27 |
| Table 5 Determination of the analysis population at Peking University Hospital of Stomatology | 28 |
| Table 6 Determination of the analysis population at Hospital of Stomatology Wuhan University | 29 |
| Table 7 Determination of the analysis population at Beijing Stomatological Hospital Capital Medical U | niversity . 30 |
| Table 8 (FAS) Analysis results of demographic data in the screening period | 31 |
| Table 9 (FAS) Analysis results of past medical history in the screening period | 32 |
| Table 9 (FAS) Analysis results of past medical history in the screening period (cont.) | 33 |
| Table 10 (FAS) Analysis results of vital signs in the preoperative examination | 34 |
| Table 11 (FAS) Analysis results of general condition as determined by the preoperative examination | ation and |
| other physical conditions | 35 |
| Table 11 (FAS) Analysis results of general condition as determined by the preoperative examination | ation and |
| other physical conditions (cont. 1) | 36 |
| Table 11 (FAS) Analysis results of general condition as determined by the preoperative examination | ation and |
| other physical conditions (cont. 2) | 37 |
| Table 12 (FAS) Analysis results of openness in the preoperative examination | 38 |
| Table 13 (FAS) Analysis results of dental examination in the preoperative examination (tooth le | vel) 39 |
| Table 13 (FAS) Analysis results of dental examination in the preoperative examination (tooth le | vel) |
| (cont. 1) | 40 |
| Table 13 (FAS) Analysis results of dental examination in the preoperative examination (tooth le | vel) |
| (cont. 2) | 41 |
| Table 13 (FAS) Analysis results of dental examination in the preoperative examination (tooth le | vel) |
| (cont. 3) | 42 |
| Table 13 (FAS) Analysis results of dental examination in the preoperative examination (tooth le | vel) |
| (cont. 4) | 43 |
| Table 13 (FAS) Analysis results of dental examination in the preoperative examination (tooth le | vel) |
| (cont. 5) | 44 |
| Table 14 (FAS) Analysis results of pregnancy test in the preoperative examination | 45 |
| Table 15 (FAS) Analysis results of oral soft tissue examination in the preoperative examination | 46 |
| Table 15 (FAS) Analysis results of oral soft tissue examination in the preoperative examination | (cont.) 47 |
| Table 16 (FAS) Analysis results of the initial screening in the preoperative examination (tooth le | evel)48 |
| Table 16 (FAS) Analysis results of the initial screening in the preoperative examination (to | |
| level) (cont.) | 49 |
| Table 17 (FAS) Analysis results of cavity preparation of diseased teeth in the screening period | 50 |
| Table 17 (FAS) Analysis results of cavity preparation of diseased teeth in the screening period ( | cont.) 51 |
| Table 18 (FAS) Analysis results of X-ray (periapical radiograph) examination before cavity pre | paration |
| in the screening period | 52 |

| $Table \ 19 \ (FAS) \ Analysis \ results \ of \ digital \ photos \ before \ cavity \ preparation \ in \ the \ screening \ period \ .$ | 53 |
|---|---|
| Table 20 (FAS) Analysis results of cavity preparation process records in the screening period | 54 |
| Table 20 (FAS) Analysis results of cavity preparation process records in the screening period (cont. | 1) 55 |
| Table 20 (FAS) Analysis results of cavity preparation process records in the screening period (cont. | <b>2</b> ) 56 |
| Table 21 (FAS) Analysis results of digital photos after cavity preparation in the screening period | 57 |
| Table 22 (FAS) Analysis results of oral soft tissue examination after cavity preparation | |
| in the screening period | 58 |
| Table 22 (FAS) Analysis results of oral soft tissue examination after cavity preparation | |
| in the screening period (cont.) | 59 |
| Table 23 (FAS) Analysis results of screening results in cavity preparation phase in the screening per | riod |
| (tooth level) | 60 |
| Table 23 (FAS) Analysis results of screening results in cavity preparation phase in the screening per | riod |
| (tooth level) (cont.) | 61 |
| Table 24 (FAS) Analysis results of intraoperative information of all diseased teeth (tooth level) | 62 |
| Table 24 (FAS) Analysis results of intraoperative information of all diseased teeth (tooth level) (con | t.) 63 |
| Table 25 (FAS) Analysis results of intraoperative records | 64 |
| Table 25 (FAS) Analysis results of intraoperative records (cont. 1) | 65 |
| Table 25 (FAS) Analysis results of intraoperative records (cont. 2) | 66 |
| Table 25 (FAS) Analysis results of intraoperative records (cont. 3) | 67 |
| Table 25 (FAS) Analysis results of intraoperative records (cont. 4) | 68 |
| Table 25 (FAS) Analysis results of intraoperative records (cont. 5) | 69 |
| $Table\ 26\ (FAS)\ Analysis\ results\ of\ digital\ photos\ taken\ immediately\ after\ the\ filling\ procedure\$ | 70 |
| Table 27 (FAS) Analysis results of oral soft tissue examination in the filling procedure | 71 |
| $Table\ 27\ (FAS)\ Analysis\ results\ of\ oral\ soft\ tissue\ examination\ during\ the\ filling\ procedure\ (cont.)$ | 72 |
| Table 28 (FAS) Analysis results of evaluation immediately after the filling procedure | 73 |
| Table 28 (FAS) Analysis results of evaluation immediately after the filling procedure (cont.) | 74 |
| Table~29~(FAS)~Analysis~results~of~consistency~evaluation~immediately~after~the~filling~procedure | 75 |
| Table 29 (FAS) Analysis results of consistency evaluation immediately after the filling | |
| procedure (cont.) | 76 |
| $Table \ 30 \ \ (FAS) \ The \ analysis \ results \ of \ primary \ efficacy \ measure - clinical \ acceptance \ rate \ of \ the \ fill$ | ling |
| at the 1 year follow-up visit after the filling procedure | 77 |
| Table 31 (FAS) The analysis results of primary efficacy measure - clinical acceptance rate of the fill | ling |
| at the 1 year follow-up visit after the filling procedure (Tipping Point analysis results) | 78 |
| Table 32 (FAS) The analysis results of primary efficacy measure - clinical acceptance rate of the fill | ling |
| at the 1 year follow-up visit after the filling procedure (subgroup analysis of each center) $\dots$ | 79 |
| Table 33 (PPS) The analysis results of primary efficacy measure - clinical acceptance rate of the filling | ing |
| at the 1 year follow-up visit after the filling procedure | 80 |
| Table 34 (PPS) The analysis results of primary efficacy measure - clinical acceptance rate of the filling | ing |
| at the 1 year follow-up visit after the filling procedure (subgroup analysis of each center) $\dots$ | 81 |
| $Table\ 35\ \ (FAS)\ The\ analysis\ results\ of\ secondary\ efficacy\ measure\ -\ clinical\ acceptance\ rate\ of\ the\ final$ | illing |
| at the 1 week follow-up visit after the filling procedure | 82 |

| Table 36 (FAS) The analysis results of secondary efficacy measures for evaluation - proximal contact, | |
|---|---|
| color match, surface roughness, surface staining, marginal discoloration, secondary caries an | d |
| pulp status 1 year after the filling procedure | 83 |
| Table 36 (FAS) The analysis results of secondary efficacy measures - proximal contact, color match, | |
| surface roughness, surface staining, marginal discoloration, secondary caries and pulp status | 1 |
| year after the filling procedure (cont.) | 85 |
| Table 37 (FAS) Analysis results of oral soft tissue examination at the 1 week ( $\pm$ 3 days) follow-up visit | |
| after the filling procedure | 86 |
| Table 37 (FAS) Analysis results of oral soft tissue examination at the 1 week (± 3 days) follow-up visit | |
| after the filling procedure (cont.) | 87 |
| Table 38 (FAS) Analysis results of filling treatment and digital photos at the 1 week (± 3 days) follow-t | ıp |
| visit after the filling procedure | 88 |
| Table 39 (FAS) Analysis results of evaluation results at the 1 week (± 3 days) follow-up visit after the | |
| filling procedure | 89 |
| Table 39 (FAS) Analysis results of evaluation results at the 1 week (± 3 days) follow-up visit after the | |
| filling procedure (cont.) | 90 |
| Table 40 (FAS) Analysis results of consistency evaluation results at the 1 week (± 3 days) follow-up vis | it |
| after the filling procedure | 91 |
| Table 42 (FAS) Analysis results of oral soft tissue examination at the 12 months (± 1 month) follow-up | |
| visit after the filling procedure | 95 |
| Table 42 (FAS) Analysis results of oral soft tissue examination at the 12 months (± 1 month) follow-up | |
| visit after the filling procedure (cont.) | 96 |
| Table 43 (FAS) Analysis results of filling treatment and digital photos at the 12 months (± 1 month) | |
| follow-up visit after the filling procedure | 97 |
| Table 44 (FAS) Analysis results of evaluation results at the 12 months (± 1 month) follow-up visit after | |
| the filling procedure | 98 |
| Table 44 (FAS) Analysis results of evaluation results at the 12 months (± 1 month) follow-up visit after | • |
| the filling procedure (cont.) | 99 |
| Table 45 (FAS) Analysis results of consistency evaluation results at the 12 months (± 1 month) follow- | пр |
| visit after the filling procedure | |
| Table 47 (FAS) Detailed descriptions of device defects | 102 |
| Table 48 (FAS) (AE) Case specific descriptions of adverse event | 103 |
| Table 49 (FAS) (AE) Summary of adverse events | 104 |
| Table 50 (FAS) Case specific descriptions of adverse events related to the investigational device | 105 |
| Table 51 (FAS) Summary of adverse events related to the investigational device | 106 |
| Table 52 (FAS) (SAE) Case specific descriptions of serious adverse events | 107 |
| Table 53 (FAS) (SAE) Summary of serious adverse events | |
| Table 54 (FAS) Case specific descriptions of serious adverse events related to the | |
| investigational device | 109 |
| Table 55 (FAS) Summary of serious adverse events related to the investigational device | 110 |
| Table 56 (FAS) List of subjects using concomitant drugs | |

#### ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviations | <b>Definitions of Terms</b> |
|---------------|-----------------------------|
| AE | Adverse Event |
| SAE | erious Adverse Event |
| FAS | Full Analysis Set |
| PPS | Per Protocol Set |
| SS | Safety Set |
| CRF | Case Report Form |

#### 1. Introduction

This document describes the specific contents of the Statistical Analysis Plan of a prospective, multi-center, randomized, controlled, and noninferiority clinical trial for the evaluation of the safety and efficacy of Filtek<sup>TM</sup> Bulk Fill Posterior Restorative in the direct restoration of Class I and II cavities of posterior teeth. When all the subjects are enrolled and complete the 1 year (±1 month) follow-up visits after the filling procedure or the trial is terminated early and the database is locked, a statistical analysis report for preoperative and 1 year (±1 month) follow-up visits after the filling procedure will be submitted for registration application. Please refer to the relevant tables, checklists, and graphs in the Statistical Analysis Plan for specific analysis items.

## 2. Background of the clinical trial

# 2.1 Background data of the disease

Composite resins for posterior restoration have been applied rapidly since the 1990s. At present, the composite resin is widely used in many countries to restore the tooth defect, contour, and function of posterior tooth in a nearly complete replacement of silver amalgam. This is mainly due to the fact that the resin has the following characteristics that the silver amalgam does not have: ① esthetic ② environmentally friendly ③ its adhesion to dental tissues is through chemical and micro-mechanical adhesion rather than simple mechanical adhesion ④ maximized preservation of healthy dental tissues. In comparison, the composite resins for posterior restoration have been greatly improved in terms of distribution, particle size, and content of filler and also mechanical and physical properties, resulting reduced polymerization shrinkage, enhanced wear resistance performance, and greatly improved clinical operational performance.

The bulk-fill material for posterior restoration (a translucent composite resin material with higher curing depth) was first applied in clinical restoration and treatment of posterior tooth defects at the start of 2000. In vitro experiments showed that the success rate of less but thicker material is the same as that

of incremental filling at a smaller thickness, while the risk of voids or failure due to thinner increment could be avoided. It is also reported in the literature that the bulk-fill materials have acceptable creep deformation, which is within the range of other composite resin materials.

3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative is a bulk-fill material. It is a filling and restoration composite material that can be activated by visible light and is optimized to restore posterior tooth more simply and quickly. When Filtek<sup>TM</sup> Bulk Fill Posterior Restorative is applied in a tooth with the methacrylate-based dental adhesive (such as the dental adhesive manufactured by 3M ESPE), the restoration can be permanently adhered to the tooth tissue. This bulk-fill resin material is more convenient and quicker to apply in comparison to the traditional composite resin materials and can save the operation time for the filling procedure.

3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative was marketed and sold in the United States, Canada, and Western Europe in September 2014 and has been widely used clinically without any AE report or complaint up to now. This trial is a pre-marketing clinical validation trial in China, and will comply the Helsinki Declaration and CFDA's Good Clinical Practice of Medical Device Clinical Trial (March 23, 2016), and will be designed and implemented in references to the requirements of CFDA's Technical Review Guidelines for the Registration of Dental Resin Filling Materials [9] and the Clinical Trial Guideline for Polymer-based Dental Restorative Materials [10] in order to evaluate the clinical safety and efficacy of Filtek<sup>TM</sup> Bulk Fill Posterior Restorative 1 week and 1 year after the restoration of Class I and II cavities of posterior teeth using a randomized controlled trial design method.

## 3. Overall design of clinical research

# 3.1 Trial objective

Evaluation of the safety and efficacy of Filtek<sup>TM</sup> Bulk Fill Posterior Restorative 1 week and 1 year after its application in the filling of Class I and II cavities of posterior teeth.

# 3.2 Selection and justification of methodology

The investigational product is a bulk-fill resin. As required in CFDA's Technical Review Guidelines for the Registration of Dental Resin Filling Materials, its clinical trial should be conducted in reference to the Clinical Trial Guideline for Polymer-based Dental Restorative Materials, which is applicable to the polymer-based dental restorative materials used in the direct restoration of posterior tooth defects, to restore Class I and II cavities of posterior teeth, in order to evaluate the safety and efficacy of 3M's Filtek<sup>TM</sup> Bulk Fill Posterior Restorative in clinical application (not including the evaluation of other new functions).

#### 3.3 Evaluation methodology of efficacy

# 1) The primary efficacy measure is the clinical acceptance rate of the filling at the 1 year follow-up visit after the filling procedure

According to the Clinical Trial Guideline for Polymer-based Dental Restorative Materials (YY/T 0990-2015), the definition of clinically acceptable filling at the 1 year follow-up visit is: grade A for retention and fracture of the filling 1 year after the filling procedure; grade A or B for marginal fracture, contour, and marginal adaptation of the filling.

#### 3.4. Secondary efficacy measures

#### 1) Clinical acceptance rate of the filling at the 1 week follow-up visit after the filling procedure:

According to the Clinical Trial Guideline for Polymer-based Dental Restorative Materials (YY/T 0990-2015), the definition of clinically acceptable filling at the 1 week follow-up is: grade A or B 1 week after the filling procedure for all the evaluation measures, including retention and fracture of the filling, marginal fracture, contour and marginal adaptation, proximal contact, color match, surface roughness, surface staining, marginal discoloration, secondary caries and pulp status;

# 2) Proximal contact, color match, surface roughness, surface staining, marginal discoloration, secondary caries and pulp status 1 year after the filling procedure

Scoring criteria for each item are listed in Appendix 1 of the protocol. The score of each item shall be recorded in the original medical record and case report form of the trial as required.

# 3.5 Evaluation methodology of safety

All AEs and SAEs will be collected and recorded from the time when the subject signs the Informed Consent to the time when the subject completes the trial or withdraws from the trial early. Primary measures include the examination of oral soft tissues and secondary caries and pulp stimulation. Because the investigational device is filling resin for posterior tooth, which will be used by local application, its safety evaluation is mainly concentrated in the oral cavity. The evaluation will be conducted before filling, immediately after filling, 1 week after filling, and 1 year after filling, in which the oral soft tissues to be examined include but not limited to buccal mucosa, lip, upper jaw, floor of mouth and tongue, and record all abnormalities and conduct statistical analysis.

The subjects can also report any local and systemic abnormalities to the investigator at any time. If necessary, they can make an appointment with the investigator for examination as soon as possible.

Evaluation methodology of secondary caries and pulp status are as stipulated in Appendix 1 of the protocol, and should be conducted before filling, immediately after filling, 1 week after filling, and 1 year after filling. If there is any abnormality and the investigator determines that it is clinically significant, it should be determined as an AE.

## 4. Investigational device/control product

#### 4.1. Investigational device

**Product name:** 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative

**Specifications and Model:** 

Kits: 4863TK, 4864TK

In syringes: 4863A1, 4863A2, 4863A3, 4863B1, 4863C2

In capsules: 4864A1, 4864A2, 4864A3, 4864B1, 4864C2

#### 4.2. Control device

**Product name:** 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT Restorative

**Specifications and Model:** 

In syringes: 7018A1B, 7018A2B, 7018A3B, 7018A3.5B, 7018B1B, 7018C2B

#### 4.3 Indications of the products

#### 4.3.1 Indications of the investigational device

- ➤ Direct restoration of anterior and posterior teeth (including occlusal surface)
- ➤ Base/liner under direct restorations
- > Core build-ups
- > Splinting
- > Indirect restorations, including inlays, onlays, and veneers
- Restorations of deciduous teeth
- Extended fissure sealing in molars and premolars
- Repair of defects in porcelain restorations, enamel, and temporaries

#### 4.3.2 Indications of the control device

- > Direct restoration of anterior and posterior teeth (including occlusal surface);
- > Post-core technique;
- Splinting;
- Indirect restorations, including inlays, onlays, and veneers.

# 5. Subject selection

#### 5.1 Inclusion criteria

- 1) Male or female, 18-70 years old (including 18 and 70 years)
- 2) Healthy, with no major systemic disease
- 3) Normal mouth openness
- 4) Molar (preferred) or premolar
- 5) Cavities satisfying any of the following 4 conditions:
  - a) Class I cavities, including those that need to be restored again after a previously failed filling;
  - b) Class II cavities, with a lesion on tooth locations other than second molars (including a failed previous filling, which needs to be filled again now), and the gingival margin after cavity preparation on the proximal surface located at the gingival crown margin;
  - c) Class II cavities, with a lesion on second molars, no missing third molars (including a failed previous filling, which needs to be filled again now), and the gingival margin after cavity preparation on the proximal surface located at the gingival crown margin;
  - d) Class II cavities, with a lesion on second molars, missing third molars, lesion on the Mesial Occlusal (MO) or Mesial Occlusal Distal (MOD) surface of second molars (including a failed previous filling, which needs to be filled again now), and the gingival margin after cavity preparation on the proximal surface located at the gingival crown margin;
- 6) Cavity size: minimum buccolingual distance on the occlusal surface (approx.) not less than 1/3 of buccolingual distance between the cusps;
- 7) The opposing tooth is natural;
- 8) Depth of the lesion reaching at least the middle layer of dentin with normal pulp vitality;
- 9) The subjects agree to participate in the trial and sign the Informed Consent;
- 10) The subject is compliant and committed to follow-up visits.

#### 5.2 Exclusion criteria

- 1) Allergic constitution or allergic to multiple drugs; allergy history of polymer based materials, such as dental resin;
- Aggressive caries; severe periodontitis; abnormal salivary gland function; temporomandibular joint disorder;
- 3) Poor oral health, DMFT: > 4 for 18~34 years old; >5 for 35~70 years old;
- 4) Teeth with special staining;
- 5) Non-carious tooth diseases, such as pathological wear (nocturnal molars, clenching habits), acid erosion, or subfissure;
- 6) Abnormal occlusion;
- 7) Severe systemic diseases; mental illness;
- 8) Breastfeeding, pregnant (positive pregnancy test result) and at childbearing age with intention to conceive;
- 9) The subject is determined to be poor compliance and could not complete the trial as required as determined by the investigator;
- 10) The cavity is determined to be unsuitable for resin filling by the investigator;
- 11) Pulp already exposed or close to be exposed at the bottom;
- 12) The subject plans to go overseas within 1 year or cannot complete the 1 year follow-up visit after the procedure due to other reasons;
- 13) The subject also participates in a clinical trial of the other drug or medical device, which has not reached its clinical endpoint;
- 14) The subject is not tolerant of or willing to use the rubber dam.

If multiple caries of a subject meet the inclusion/exclusion criteria, the investigator will select the enrolled tooth by giving priority to molars; If all the teeth that meet the inclusion/exclusion criteria are molars, the investigator can enroll any tooth and indicate the enrolled tooth number in the original medical record and case report form. If other teeth that are not included need to be treated at the same

time, the name of filling resin (when other marketed products than Filtek<sup>TM</sup> Z350XT are required) and the tooth location number for such filling should be recorded.

#### 6. General statistical considerations

#### 6.1 Determination of the sample size and its justifications

#### **6.1.1 Statistical design (Test of Hypothesis)**

This trial will adopt a prospective, multicenter, randomized, and controlled design, using the Filtek<sup>TM</sup> Z350XT as the control, which is also a resin filling material and has similar and comparable characteristics, uses, and indications to the investigational device. The noninferiority design will be adopted to prove that the safety and efficacy of the investigational device are not inferior to the control device, which was already approved for marketing with clinically validated safety and efficacy. Corresponding statistical design and test of hypothesis are:

$$\mathbf{H}_0: p_T - p_C \le -\Delta$$

$$\mathbf{H}_1: p_T - p_C \ge -\Delta$$

Where  $p_T$  is the expected success rate of the filling in corresponding treatment group,  $p_C$  is the expected success rate of the control group and  $\Delta$  is the noninferiority margin (absolute value).

# **6.1.2** Total sample size

It is estimated that 240 patients will be enrolled in this trial, and randomly assigned to the treatment or control group at 1:1 ratio. The number of cases in each group is 120. The calculation of the sample size is based on the primary endpoint measure, i.e. clinical acceptance rate of the filling at the 1 year follow-up visit.

Since the scope of application of the investigational device is direct or indirect restoration of both anterior and posterior teeth, and based on existing clinical evidence and estimation by the clinical experience of experts, and assuming the clinical acceptance rate in the control group 1 year after treatment is 97% and it is estimated that the treatment group can reach the same effective level after using the investigational product, with a clinically recognized noninferiority margin of 7% after discussion, a significance level of 5% at two tails, a statistical power of 80%, and a maximum possible dropout rate of 20%, about 120 patients should be included in each group with a total of 240 patients to be included in both groups.

Corresponding sample size calculation is:

$$n = \frac{\left[\mu_{1-\alpha} \sqrt{2 \,\overline{p}(1-\overline{p})} + \mu_{1-\beta} \sqrt{p_T(1-p_T) + p_C(1-p_C)}\right]^2}{\left(\Delta - (p_T - p_C)\right)^2}$$

Where  $p_T$  is the expected fusion effectiveness of the treatment group,  $p_C$  is the expected effectiveness of the control group,  $p_C$  is the mean effectiveness of both groups,  $p_C$  is the noninferiority margin,  $p_C$  is the quantile of standard normal distribution,  $p_C$  is the level of Type I Error, which is set at 0.025, and  $p_C$  is the level of Type II Error, which is set at 0.2.

#### 6.2 Analysis population

- 1) Safety Set (SS): include all the subjects who are enrolled, receive the filling, and complete at least 1 follow-up visit.
- 2) Full analysis set (FAS): the set of subjects determined according to the Intention-To-Treat principle, which refers to the data set composed of all the subjects who are included in randomization and receive the investigational product.
- 3) Per Protocol Set (PPS): refers to the subgroup of treatment population who are included in randomization and receive the investigational product, while excluding those who seriously violate the protocol (referring to the violation of the inclusion criteria or exclusion criteria by the subjects, etc.).

The analysis of primary efficacy measures will be based on the FAS and PPS at the same time. In addition, all baseline demographic data and analysis of secondary efficacy measures will be based on the FAS, so as to the safety evaluation (SS is the same as FAS in terms of definitions, and thus is not defined separately).

#### 6.3 Determination rules and flow diagram of analysis population data set

- (1) No investigational device is used: the subject is assigned a random number, but does not receive any trial related treatment (treatment group, control group, or a third-party product);
- (2) Violation of the inclusion and exclusion criteria: the subject does not meet the inclusion criteria or meets the exclusion criteria defined by the protocol, and their violation of the protocol will seriously affect the evaluation results of primary efficacy measures; such violations will be determined jointly by the sponsor, investigators, and biometrician on whether they seriously affect the evaluation results of the primary efficacy measures via discussion in the peer review meetings;
- (3) Lost to follow-up in the trial: the primary endpoint measure of a subject clinical acceptance rate of the filling at the 1 year follow-up visit after the filling procedure cannot be acquired.
- (4) Cross assignment: The subjects randomly assigned to the treatment group use the product for the control group, and vice versa;
- (5) Use of an investigational product out of spec: the specifications of the device used by the subject is not within the range specified in the protocol;
- (6) Use of a third-party product: the subject who is randomly assigned to the treatment or control group receives a third-party product;
- (7) FAS = number of randomly assigned subjects number of subjects who do not receive any investigational device;

PPS = FAS - number of subjects who are in serious deviation to the protocol;

Number of subjects who are in serious deviation to the protocol = number of subjects who fail inclusion and exclusion criteria + number of subjects who are lost to follow-up in the trial + number of subjects who are crossly assigned + number of subjects who receive an out of spec investigational product + number of subjects who receive a third party product;

Priorities of deviations to the protocol are: lost to follow-up in the trial; cross assignment; use of a third party product; use of an out of spec product; failing inclusion and exclusion criteria. If a subject satisfies two or more above violations, they will be categorized by the aforesaid priority;

All deviations to the protocol in tabulated statistical analysis will be listed depending on actual situations. If the number of subjects who receive out of spec products is 0, it cannot be displayed in the table. At the same time, the subjects who do not receive any investigational device or are in serious deviation to the protocol will be listed, including the center code, randomization number, group, gender, age, type, reason, FAS, and PPS.



Fig. 1 Determination flow diagram of analysis population data set

#### 6.4 Missing values, abnormal values, and outliers

For the analysis of possible missing data in the process, Carry Forward methods will be used for missing data of primary efficacy measures in principle. For the primary endpoint measures, CMH Chi square test adjusted for center effect will be used for estimating the difference between two groups on clinical acceptance rate and its 95% Confidence Interval. In above analyses, the Worst Case Carry Forward (WCCF) and Last Observation Carried Forward (LOCF) approaches will be used to carry forward the missing data of primary endpoint measures. For the missing data of other measures, Carry Forward strategy will not be applied, while actual observation data will be analyzed directly.

Wrong and unreasonable data will be handled in the data cleaning process before statistical analysis. The information of patients, who withdraw or are removed from the trial, will be included in the final statistical analysis. In the Statistical Report, specific reasons for all withdrawals or removals will be described in detail, while those missing primary measures due to early withdrawal will be analyzed according to the aforesaid missing value handling strategy.

#### 6.5 Significance level and statistical analysis software

For primary endpoint measures, a significance level of 0.025 at one tail (corresponding to one side 95% CI) will be set for all statistical analyses. For other measures, all statistical analyses will be performed a significance level of 0.05 at two tails (except for those are specially noted). All statistical analyses will be performed using the statistical software SAS® 9.4.

#### 6.6 Consolidation of centers

This trial will be carried out in several clinical trial institutions at the same time, and the actual numbers of successful enrolled subjects in each center will be different. In order to avoid the impact of small sample size in each center on stability and reliability of the analysis results of primary endpoints, the centers where less than 10 subjects are successful enrolled will be consolidated. Based on past experience and reference, the following two methods will be generally adopted for the consolidation of centers:

- (1) The centers with the number of actually enrolled subjects < 10 will be sorted by the center code and then directly consolidated until the number of consolidated subjects is  $\ge 10$ ;
- (2) The centers will be consolidated based on adjacency, and the number of consolidated subjects should be  $\geq 10$ ;

Analysis methods for the consolidation of centers in statistical analysis will be determined jointly by the sponsor, investigators, and biometrician via discussion in the peer review meetings.

#### 7. Statistical analysis measures and methodology

#### 7.1 Demographic data and other baseline data

Demographic data include age, sex, and clinical diagnosis. Other baseline data include previous medical history, vital signs, general condition as determined by preoperative examination and other physical conditions, openness, dental examination, pregnancy test, oral soft tissue examination, preoperative preliminary screening results, cavity preparation of diseased teeth, whether to perform X-ray periapical radiograph before cavity preparation, digital photos taken before cavity preparation, records of cavity preparation process, digital photo taken after cavity preparation, oral soft tissue examination after cavity preparation, screening results in cavity preparation phase and other relevant measures.

Where,

Age = (Date of Informed Consent - Date of Birth) /365.25;

These measures are mainly descriptive information. Count data will be described by frequency and constituent ratio. Measurement data will be described by mean value, standard deviation, median, interquartile range, maximum, and minimum. Likelihood  $\chi 2$  test will be used for group comparison of the count data, while Fisher's exact test will be used when the theoretical frequency is lower than 5 in more than 25% cells. For group comparison of measurement data, group t-test will be used for those that are normally distributed, while Wilcoxon Rank Sum test will be used for those that are not normally distributed.

# 7.2 Operation information

The intraoperative information includes the information of all diseased teeth recorded during the operation, intraoperative records, digital photos taken immediately after the filling procedure, oral soft tissue examination during the filling procedure, immediate evaluation after the filling procedure, and other relevant measures.

These measures are mainly descriptive information. Their statistical analysis methodology is the same as those in 7.1.

# 7.3 Primary efficacy measures

Clinical acceptance rate of the filling at the 1 year follow-up visit after the filling procedure Calculation:

According to the Clinical Trial Guideline for Polymer-based Dental Restorative Materials (YY/T 0990-2015), the definition of clinically acceptable filling at the 1 year follow-up visit is: grade

A for retention and fracture of the filling 1 year after the filling procedure; grade A or B for marginal fracture, contour, and marginal adaptation of the filling.

- 1) For the "retention and fracture", "marginal fracture", and "contour and marginal adaptation", if any of the above measures is void or NA, the clinical acceptance is "Void";
- 2 If the "retention and fracture" is scored as A and "marginal fracture" and "contour and marginal adaptation" are scored as A or B, the clinical acceptance is "Yes";
- 3 If the "retention and fracture" is scored as B or C, or "marginal fracture" is scored as C, or "contour and marginal adaptation" is scored as C, the clinical acceptance is "No";

For the primary efficacy measure, CMH Chi square test adjusted for center effect will be used for group comparison, and the difference between groups on efficacy and its 95% CI will also be estimated. If the 95% CI of the difference between groups on efficacy is greater than -7%, the investigational product is deemed as not inferior to the control product. Meanwhile, the clinical acceptance rate and its 95% CI estimated by Tipping Point (Cut-off value approach) will be used as the results of the sensitivity analysis.

If the trial results show that there are significant differences between the treatment and control groups on other baseline variables (such as age, sex, etc.), these situations will be fully communicated with the investigators in the data analysis phase. Based on one way analysis results of baseline variables and primary endpoint measures, previous literature references and the experiences of clinical experts, unbalanced measures between groups that affected the primary end points, namely, confounding factors, will be further clarified. These factors will be considered to be put into the generalized linear model for correction, as the sensitivity analysis of the primary endpoint measure.

## 7.4. Secondary efficacy measures

# (1) Clinical acceptance rate of the filling at the 1 week follow-up visit after the filling procedure Calculation:

According to the Clinical Trial Guideline for Polymer-based Dental Restorative Materials (YY/T 0990-2015), the definition of clinically acceptable filling at the 1 week follow-up is: grade A or B 1 week after the filling procedure for all the evaluation measures, including retention and fracture of the filling, marginal fracture, contour and marginal adaptation, proximal contact, color match, surface roughness, surface staining, marginal discoloration, secondary caries and pulp status;

① In all of the measures 1 week after the filling procedure, including retention and fracture, marginal fracture, contour and marginal adaptation, proximal contact, color match, surface roughness,

surface staining, marginal discoloration, secondary caries and pulp status, if any of above measures is void or NA, the clinical acceptance is "Void";

- 2 If all the measures 1 week after the filling procedure, including retention and fracture, marginal fracture, contour and marginal adaptation, proximal contact, color match, surface roughness, surface staining, marginal discoloration, secondary caries and pulp status, are scored as A or B, the clinical acceptance is "Yes";
- ③ If all the measures 1 week after the filling procedure, including retention and fracture, marginal fracture, contour and marginal adaptation, proximal contact, color match, surface roughness, surface staining, marginal discoloration, secondary caries and pulp status, are scored not as those in ① or ②, the clinical acceptance is "No";

# (2) Proximal contact, color match, surface roughness, surface staining, marginal discoloration, secondary caries and pulp status 1 year after the filling procedure

These measures will be analyzed based on actual data and are mainly descriptive information. Their statistical analysis methodology is the same as those in 7.1.

# 7.5 Safety measures

- (1) Incidence of SAEs (Serious Adverse Events)
- (2) Incidence of AEs (Adverse Events)

This section will provide the incidences of AEs and SAEs and the results of group comparison analysis. Their statistical analysis methodology is the same as those in 7.1.

# 7.6 Follow-up data

Follow-up data include data from oral soft tissue examination, filling treatment, digital photos, evaluation of follow-up measures, and other measures. The follow-up time points include 1 week ( $\pm$  3 days) after the filling procedure and 12 months ( $\pm$  1 month) after the filling procedure.

Descriptive analysis will be mainly used for the relevant measures of follow-up data.

# 7.7 X-ray examination

For X-ray examination measure, the results of descriptive analysis will be provided, i.e., whether X-ray (periapical radiograph) examination is performed immediately, at the 1 week ( $\pm$  3 days) and 12 months ( $\pm$  1 month) follow-up visit after the filling procedure, and whether X-ray examination results are abnormal. In addition, the outcomes immediately after the filling procedure, at the 1 week ( $\pm$  3 days)

and 12 months ( $\pm$  1 month) follow-up visit after the filling procedure in comparison to the screening period will also be provided, including four situations: "Normal  $\rightarrow$  Abnormal", "Normal  $\rightarrow$  Normal", "Abnormal  $\rightarrow$  Normal", and "Abnormal  $\rightarrow$  Abnormal", mainly using the descriptive analysis methods.

#### 7.8 Device defects

Device defects will be presented in a list. List specific descriptions of device defects for subjects will include the center code, randomization number, group assignment, age, gender, applicable items to a device defect, attribution of the device defect, number, name of the device defect, starting time, ending time, details of the device defect, results of the device defect, measures taken, any resulting medical events, diseases, or injuries, whether to return to the sponsor and other measures.

#### 7.9 AEs and SAEs

AEs and those related to the investigational device will be provided by a list and summary of subjects. The list of subjects for AEs and those related to the investigational device will include the center code, randomization number, group assignment, gender, age, name of AE, occurrence time (days) after the procedure, remission time (days), characteristics of AE, number of paroxysmal attacks, severity, record and report of AEs, relationship to the investigational device, outcomes, sequela, corrective treatment, withdrawal, SAEs, and other measures.

Where the AEs related to the investigational device refer to AEs that are "possibly related" or "quite possibly related" or "definitely related" to the investigational device.

Occurrence time after the procedure (days) = starting date of AE - date of cavity filling,

Remission time (days) = ending date of AE - starting date of AE.

The summary table will list the total number of AEs/those related to the investigational device, and the total cases of all AEs/those related to the investigational device.

Where the total cases of AEs refer to the number of subjects with AEs. A subject with one occurrence of AE will be deemed as "Yes";

SAEs and those related to the investigational device will be provided by a list and summary of subjects. The list of subjects for SAEs and those related to the investigational device will include the center code, randomization number, group assignment, gender, age, name of SAE, occurrence time (days) after the procedure, remission time (days), characteristics of SAE, number of paroxysmal attacks, severity, relationship to the investigational device, outcomes, sequela, corrective treatment, withdrawal, report type, SAE situations, and reports.

Where the calculation of occurrence time after the procedure (days) and remission time (days), summary table format, and statistical principles are the same as those for AEs.

#### 7.10 Concomitant medication

Concomitant drugs will be presented in a list. List of subjects for concomitant drugs include the center code, randomization number, group assignment, age, gender, drug name, whether still in use, administration route, dosage, unit, indications, and treatment reasons.

## 8. GENERATION OF STATISTICAL TABLES, LISTS, AND GRAPHS



Fig. 1 Determination flow diagram of the analysis population data set

Table 1 Determination of the analysis population

| asures | Treatment group | Control group |
|---|---|---|
| Random assignment | XXX (XX.X%) | XXX (XX.X%) |
| Subjects who do not receive any investigational device | XXX (XX.X%) | XXX (XX.X%) |
| Serious deviation to the protocol | | |
| Failing inclusion and exclusion criteria | XXX (XX.X%) | XXX (XX.X%) |
| Lost to follow-up | XXX (XX.X%) | XXX (XX.X%) |
| Cross assignment | XXX (XX.X%) | XXX (XX.X%) |
| Use of a third party product | XXX (XX.X%) | XXX (XX.X%) |
| Use of an investigational product out of spec | XXX (XX.X%) | XXX (XX.X%) |
| FAS | XXX (XX.X%) | XXX (XX.X%) |
| PPS | XXX (XX.X%) | XXX (XX.X%) |

- Notes: 1: FAS = number of randomly assigned subjects number of subjects who do not receive any investigational device;
  - PPS = FAS number of subjects who are in serious deviation to the protocol;
  - 2: No investigational device is used: the subject is assigned a random number, but does not receive any trial related treatment;
    - Lost to follow-up in the trial: the primary endpoint measure of a subject clinical acceptance rate at the 1 year follow-up visit after the filling procedure cannot be acquired.
    - Failing inclusion and exclusion criteria: the subject does not meet the inclusion criteria or meets the exclusion criteria defined by the protocol;
    - Use of an investigational product out of spec: the specifications of the device used by the subject is not within the range specified in the protocol;
    - Cross assignment: The subjects randomly assigned to the treatment group use the product for the control group, and vice versa;
    - Use of a third-party product: the subject who is randomly assigned to the treatment or control group receives a third-party product;
  - 3: Number of subjects who are in serious deviation to the protocol = number of subjects who fail inclusion and exclusion criteria + number of subjects who are lost to follow-up in the trial + number of subjects who are crossly assigned + number of subjects who receive a third party product + number of subjects who receive an out of spec investigational product;
  - 4: Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 2 List of subjects who do not receive any investigational device or are in serious deviation to the protocol

| Center code | Randomization No. | Group | Sex | Age | Type | Reason | FAS | PPS |
|---|---|---|---|---|---|---|---|---|
| XXX<br>XXX | XXX<br>XXX | XXX<br>XXX | XXX<br>XXX | XXX<br>XXX | • • • • • | | | |

Notes: fill out a "\" for subjects included in SS and FAS (PPS) analysis and an "x" if not.

Table 3 Statistical analysis results of subjects in serious deviation to the protocol (CRF collection)

| Measures | Treatment group | Control group |
|---|---|---|
| Group assignment | XXX <sup>#1</sup> (XXX <sup>#2</sup> ) | XXX (XXX) |
| Informed Consent process not followed | $XXX (XX^{#2}, XX.X\%^{#3})$ | XXX (XX, XX.X%) |
| Failing inclusion/exclusion criteria | XXX (XX, XX.X%) | XXX (XX, XX.X%) |
| Procedures/steps not in compliance with the protocol | XXX (XX, XX.X%) | XXX (XX, XX.X%) |
| Procedures/steps omitted | XXX (XX, XX.X%) | XXX (XX, XX.X%) |
| A certain visit is omitted | XXX (XX, XX.X%) | XXX (XX, XX.X%) |
| Record/report of AEs not as required | XXX (XX, XX.X%) | XXX (XX, XX.X%) |
| Use of investigational or control device not by Instruction for Use | XXX (XX, XX.X%) | XXX (XX, XX.X%) |
| Clinical visits required by the protocol are not in specified time window | XXX (XX, XX.X%) | XXX (XX, XX.X%) |
| Storage of investigational/control device not as required | XXX (XX, XX.X%) | XXX (XX, XX.X%) |
| Other | XXX (XX, XX.X%) | XXX (XX, XX.X%) |

Notes: 1. #1: Total number of deviations to the protocol

<sup>#2:</sup> Total cases of deviations to the protocol

<sup>#3:</sup> Percentage = total number of a deviation/total cases of deviations to the protocol\*100%.

Table 4 List of subjects in serious deviation to the protocol (CRF collection)

| Center<br>code | Randomization<br>No. | · | | Age | Follow-<br>up visit<br>time<br>window | Type | Details of deviations<br>to the protocol | | SS | FAS | PPS |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX | XXX | | | | XXX | | XXX | XXX | XXX | XXX | XXX |
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Table 5 Determination of the analysis population at Peking University Hospital of Stomatology

| Measures | Treatment group | Control group |
|---|---|---|
| Random assignment | XXX (XX.X%) | XXX (XX.X%) |
| Subjects who do not receive any investigational device | XXX (XX.X%) | XXX (XX.X%) |
| Serious deviation to the protocol | | |
| Failing inclusion and exclusion criteria | XXX (XX.X%) | XXX (XX.X%) |
| Lost to follow-up | XXX (XX.X%) | XXX (XX.X%) |
| Cross assignment | XXX (XX.X%) | XXX (XX.X%) |
| Use of a third party product | XXX (XX.X%) | XXX (XX.X%) |
| Use of an investigational product out of spec | XXX (XX.X%) | XXX (XX.X%) |
| FAS | XXX (XX.X%) | XXX (XX.X%) |
| PPS | XXX (XX.X%) | XXX (XX.X%) |

- Notes: 1: FAS = number of randomly assigned subjects number of subjects who do not receive any investigational device;
  - PPS = FAS number of subjects who are in serious deviation to the protocol;
  - 2: No investigational device is used: the subject is assigned a random number, but does not receive any trial related treatment;
    - Lost to follow-up in the trial: the primary endpoint measure of a subject clinical acceptance rate at the 1 year follow-up visit after the filling procedure cannot be acquired.
    - Failing inclusion and exclusion criteria: the subject does not meet the inclusion criteria or meets the exclusion criteria defined by the protocol;
    - Use of an investigational product out of spec: the specifications of the device used by the subject is not within the range specified in the protocol;
    - Cross assignment: The subjects randomly assigned to the treatment group use the product for the control group, and vice versa;
    - Use of a third-party product: the subject who is randomly assigned to the treatment or control group receives a third-party product;
  - 3: Number of subjects who are in serious deviation to the protocol = number of subjects who fail inclusion and exclusion criteria + number of subjects who are lost to follow-up in the trial + number of subjects who are crossly assigned + number of subjects who receive a third party product + number of subjects who receive an out of spec investigational product;
  - 4: Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 6 Determination of the analysis population at Hospital of Stomatology Wuhan University

| Measures . | Treatment group | Control group |
|---|---|---|
| Random assignment | XXX (XX.X%) | XXX (XX.X%) |
| Subjects who do not receive any investigational device | XXX (XX.X%) | XXX (XX.X%) |
| Serious deviation to the protocol | ` , | , , |
| Failing inclusion and exclusion criteria | XXX (XX.X%) | XXX (XX.X%) |
| Lost to follow-up | XXX (XX.X%) | XXX (XX.X%) |
| Cross assignment | XXX (XX.X%) | XXX (XX.X%) |
| Use of a third party product | XXX (XX.X%) | XXX (XX.X%) |
| Use of an investigational product out of spec | XXX (XX.X%) | XXX (XX.X%) |
| FAS | XXX (XX.X%) | XXX (XX.X%) |
| PPS | XXX (XX.X%) | XXX (XX.X%) |

- Notes: 1: FAS = number of randomly assigned subjects number of subjects who do not receive any investigational device;
  - PPS = FAS number of subjects who are in serious deviation to the protocol;
  - 2: No investigational device is used: the subject is assigned a random number, but does not receive any trial related treatment;
    - Lost to follow-up in the trial: the primary endpoint measure of a subject clinical acceptance rate at the 1 year follow-up visit after the filling procedure cannot be acquired.
    - Failing inclusion and exclusion criteria: the subject does not meet the inclusion criteria or meets the exclusion criteria defined by the protocol;
    - Use of an investigational product out of spec: the specifications of the device used by the subject is not within the range specified in the protocol;
    - Cross assignment: The subjects randomly assigned to the treatment group use the product for the control group, and vice versa;
    - Use of a third-party product: the subject who is randomly assigned to the treatment or control group receives a third-party product;
  - 3: Number of subjects who are in serious deviation to the protocol = number of subjects who fail inclusion and exclusion criteria + number of subjects who are lost to follow-up in the trial + number of subjects who are crossly assigned + number of subjects who receive a third party product + number of subjects who receive an out of spec investigational product;
  - 4: Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 7 Determination of the analysis population at Beijing Stomatological Hospital Capital Medical University

| Measures | Treatment group Control grou | |
|---|---|---|
| Random assignment | XXX (XX.X%) | XXX (XX.X%) |
| Subjects who do not receive any investigational device | XXX (XX.X%) | XXX (XX.X%) |
| Serious deviation to the protocol | | |
| Failing inclusion and exclusion criteria | XXX (XX.X%) | XXX (XX.X%) |
| Lost to follow-up | XXX (XX.X%) | XXX (XX.X%) |
| Cross assignment | XXX (XX.X%) | XXX (XX.X%) |
| Use of a third party product | XXX (XX.X%) | XXX (XX.X%) |
| Use of an investigational product out of spec | XXX (XX.X%) | XXX (XX.X%) |
| FAS | XXX (XX.X%) | XXX (XX.X%) |
| PPS | XXX (XX.X%) | XXX (XX.X%) |

- Notes: 1: FAS = number of randomly assigned subjects number of subjects who do not receive any investigational device;
  - PPS = FAS number of subjects who are in serious deviation to the protocol;
  - 2: No investigational device is used: the subject is assigned a random number, but does not receive any trial related treatment;
    - Lost to follow-up in the trial: the primary endpoint measure of a subject clinical acceptance rate at the 1 year follow-up visit after the filling procedure cannot be acquired.
    - Failing inclusion and exclusion criteria: the subject does not meet the inclusion criteria or meets the exclusion criteria defined by the protocol;
    - Use of an investigational product out of spec: the specifications of the device used by the subject is not within the range specified in the protocol;
    - Cross assignment: The subjects randomly assigned to the treatment group use the product for the control group, and vice versa;
    - Use of a third-party product: the subject who is randomly assigned to the treatment or control group receives a third-party product;
  - 3: Number of subjects who are in serious deviation to the protocol = number of subjects who fail inclusion and exclusion criteria + number of subjects who are lost to follow-up in the trial + number of subjects who are crossly assigned + number of subjects who receive a third party product + number of subjects who receive an out of spec investigational product;
  - 4: Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 8 (FAS) Analysis results of demographic data in the screening period

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Age (yr) | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | XX. $XX \pm XX$ . $XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Sex | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Male | XXX (XX.X%) | XXX (XX.X%) | | |
| Female | XXX (XX.X%) | XXX (XX.X%) | | |
| Clinically diagnosed caries | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| None | XXX (XX.X%) | XXX (XX.X%) | | |
| With | XXX (XX.X%) | XXX (XX.X%) | | |
| Clinically diagnosed other | , , | , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| None | XXX (XX.X%) | XXX (XX.X%) | | |
| With | XXX (XX.X%) | XXX (XX.X%) | | |

- Notes: 1. Likelihood  $\chi^2$  test or Fisher's exact probability test will be used for group comparison of qualitative measures.
  - 2. Group t-test or Wilcoxon Rank Sum test will be used for group comparison of quantitative measures.
  - 3. For quantitative measures Q1: 25th quantile Q3: 75th quantile.
  - 4. Age = (Date of Informed Consent Date of Birth)/365.25;
  - 5. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

31 / 111

Table 9 (FAS) Analysis results of past medical history in the screening period

| Measures | | Control group | Statistics | P value |
|---|---|---|---|---|
| Smoking history | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Never | XXX (XX.X%) | XXX (XX.X%) | | |
| Still | XXX (XX.X%) | XXX (XX.X%) | | |
| Quit | XXX (XX.X%) | XXX (XX.X%) | | |
| Smoking history Still Years of sm | oking | , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Smoking history Still Number of | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean ± SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Smoking history Quit Years of sm | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Smoking history Quit Years of qu | 2 | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Allergy history | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| None | XXX (XX.X%) | XXX (XX.X%) | | |
| With | XXX (XX.X%) | XXX (XX.X%) | | |
| Subject had a dental history prior to | enrollment | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| None | XXX (XX.X%) | XXX (XX.X%) | | |
| With | XXX (XX.X%) | XXX (XX.X%) | | |
| Had dental history Currently taking | medication | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Had dental history Cured or not | . , | , , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures. 2. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 9 (FAS) Analysis results of past medical history in the screening period (cont.)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| History of other diseases | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| None | XXX (XX.X%) | XXX (XX.X%) | | |
| With | XXX (XX.X%) | XXX (XX.X%) | | |
| History of other diseases | , , | , , | | |
| Currently taking medication | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| History of other diseases | · | · · · · · | | |
| Cured or not | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures. 2. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 10 (FAS) Analysis results of vital signs in the preoperative examination

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Systolic (mmHg) | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Diastolic (mmHg) | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean $\pm$ SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Heart rate (beats/minute) | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX. XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Respiration rate (times/minute) | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean ± SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |

- Notes: 1. Group t-test or Wilcoxon Rank Sum test will be used for group comparison of quantitative measures.
  - 2. For quantitative measures Q1: 25th quantile Q3: 75th quantile.
  - 3. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 11 (FAS) Analysis results of general condition as determined by the preoperative examination and other physical conditions

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| General condition | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Very good | XXX (XX.X%) | XXX (XX.X%) | | |
| Good | XXX (XX.X%) | XXX (XX.X%) | | |
| General | XXX (XX.X%) | XXX (XX.X%) | | |
| Poor | XXX (XX.X%) | XXX (XX.X%) | | |
| Very poor | XXX (XX.X%) | XXX (XX.X%) | | |
| Heart disease | , | , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| None | XXX (XX.X%) | XXX (XX.X%) | | |
| With | XXX (XX.X%) | XXX (XX.X%) | | |
| Heart disease Coronary disease | 11111 (1111117,0) | 11111 (11111173) | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | 71.721.71 | 71.77.171 |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Heart disease Hypertension | 71111 (11111170) | 71111 (7111117 o) | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | 71.71717171 | 71.71717171 |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Heart disease Arrhythmia | 71711 (7171.7170) | 71.71 (71.71.70) | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | 71.71.71.71 | 21.222221 |
| Yes | XXX(XX.X%) | XXX (XX.X%) | | |
| Heart disease Other | AAA(AA.A70) | $\mathcal{M}\mathcal{M}(\mathcal{M}\mathcal{M},\mathcal{M}/0)$ | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XXX)<br>XXX (XX.X%) | Λ.ΛΛΛΛ | Α.ΑΑΑΑ |
| Yes | XXX(XX.X%) | XXX (XX.X%) | | |
| Respiratory diseases | $\Lambda\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda/0)$ | $\Lambda\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda/0)$ | | |
| Cases (Nmiss) | XXX (XXX) | VVV (VVV) | X.XXXX | X.XXXX |
| None | XXX (XXX)<br>XXX (XX.X%) | XXX (XXX)<br>XXX (XX.X%) | Λ.ΛΛΛΛ | Λ.ΛΛΛΛ |
| With | XXX (XX.X%) | XXX (XX.X%) | | |
| Respiratory diseases Cough | $\Lambda\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda/0)$ | $\Lambda\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda/0)$ | | |
| Cases (Nmiss) | VVV (VVV) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XXX)<br>XXX (XX.X%) | XXX (XX.X%) | Λ.ΛΛΛΛ | Λ.ΛΛΛΛ |
| | | ` , | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Respiratory diseases Asthma | VVV (VVV) | VVV (VVV) | VVVVV | v vvvv |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Respiratory diseases Pneumonia | 7/7/7/ (3/7/7/) | 7777 (7777) | 37 37373737 | 37 37373737 |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |

Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures.

 $<sup>2. \</sup> Treatment \ group: 3M^{TM} \ Filtek^{TM} \ Bulk \ Fill \ Posterior \ Restorative; Control \ group: 3M^{TM} \ Filtek^{TM} \ Z350XT.$ 

Table 11 (FAS) Analysis results of general condition as determined by the preoperative examination and other physical conditions (cont. 1)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Respiratory diseases Bronchitis | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Respiratory diseases Other | , | , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Infectious diseases | , | , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| None | XXX (XX.X%) | XXX (XX.X%) | | |
| With | XXX (XX.X%) | XXX (XX.X%) | | |
| Infectious diseases Hepatitis | () | ( | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | 1111111111 | 1111111111 |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Infectious diseases HBsAg positive | | 11111 (111111170) | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | 71 | 11.71.71.71 |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Infectious diseases Tuberculosis | 71.71 (71.71.70) | 717171 (7171.7170) | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | 71.72727 | 71.71.71.71 |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Infectious diseases AIDS | $\Lambda\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda/0)$ | $\Lambda\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda/0)$ | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XXX)<br>XXX (XX.X%) | XXX (XXX)<br>XXX (XX.X%) | Α.ΑΑΑΑ | Λ.ΛΛΛΛ |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Infectious diseases Other | $\Lambda\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda/0)$ | $\Lambda\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda/0)$ | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XXX)<br>XXX (XX.X%) | Λ.ΛΛΛΛ | Λ.ΛΛΛΛ |
| Yes | XXX (XX.X%) | | | |
| Other conditions Diabetes | $\Lambda\Lambda\Lambda$ ( $\Lambda\Lambda.\Lambda$ 70) | XXX (XX.X%) | | |
| | VVV (VVV) | VVV (VVV) | X.XXXX | X.XXXX |
| Cases (Nmiss)<br>No | XXX (XXX) | XXX (XXX) | Λ.ΛΛΛΛ | Λ.ΛΛΛΛ |
| | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Other conditions Nephrosis | VVV (VVV) | VVV (VVV) | VVVVV | vvvvv |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Other conditions Rheumatism | WWW (WWW) | VVV (VVV) | 3/ 3/3/3/3/ | 3/ 3/3/3/3/ |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |

Notes: 1. Likelihood  $\chi^2$  test or Fisher's exact probability test will be used for group comparison of qualitative measures.

<sup>2.</sup> Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.
Table 11 (FAS) Analysis results of general condition as determined by the preoperative examination and other physical conditions (cont. 2)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Other conditions Mental illne | ess | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Other conditions Epilepsy/co | nvulsion | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Other conditions Fever | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Other conditions Hemorrhagia | ic tendency | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Other conditions Malignant t | umor | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Other conditions Regurgitation | on and belching | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Other conditions Other | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | ` / | | |
| Yes | XXX (XX.X%) | | | |

Notes: 1. Likelihood  $\chi^2$  test or Fisher's exact probability test will be used for group comparison of qualitative measures.

<sup>2.</sup> Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 12 (FAS) Analysis results of openness in the preoperative examination

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Openness | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| Limited | XXX (XX.X%) | XXX (XX.X%) | | |
| If limited, the width of openness (cm) | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |

- Notes: 1. Likelihood  $\chi^2$  test or Fisher's exact probability test will be used for group comparison of qualitative measures.
  - 2. Group t-test or Wilcoxon Rank Sum test will be used for group comparison of quantitative measures.

    3. For quantitative measures Q1: 25th quantile Q3: 75th quantile.

  - 4. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 13 (FAS) Analysis results of dental examination in the preoperative examination (tooth level)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Dental examination (subject level) | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Done | XXX (XX.X%) | XXX (XX.X%) | | |
| Not done | XXX (XX.X%) | XXX (XX.X%) | | |
| Caries (subject level) | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| None | XXX (XX.X%) | XXX (XX.X%) | | |
| With | XXX (XX.X%) | XXX (XX.X%) | | |
| Number of caries (subject level) | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 1 | XXX (XX.X%) | XXX (XX.X%) | | |
| 2 | XXX (XX.X%) | XXX (XX.X%) | | |
| | XXX (XX.X%) | XXX (XX.X%) | | |
| Location of caries | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| UR | XXX (XX.X%) | XXX (XX.X%) | | |
| UL | XXX (XX.X%) | XXX (XX.X%) | | |
| LL | XXX (XX.X%) | XXX (XX.X%) | | |
| LR | XXX (XX.X%) | XXX (XX.X%) | | |
| Code of UR caries | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 11 | XXX (XX.X%) | XXX (XX.X%) | | |
| 12 | XXX (XX.X%) | XXX (XX.X%) | | |
| 13 | XXX (XX.X%) | XXX (XX.X%) | | |
| 14 | XXX (XX.X%) | XXX (XX.X%) | | |
| 15 | XXX (XX.X%) | XXX (XX.X%) | | |
| 16 | XXX (XX.X%) | XXX (XX.X%) | | |
| 17 | XXX (XX.X%) | XXX (XX.X%) | | |
| 18 | XXX (XX.X%) | XXX (XX.X%) | | |
| Code of UL caries | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 21 | XXX (XX.X%) | XXX (XX.X%) | | |
| 22 | XXX (XX.X%) | XXX (XX.X%) | | |
| 23 | XXX (XX.X%) | XXX (XX.X%) | | |
| 24 | XXX (XX.X%) | XXX (XX.X%) | | |
| 25 | XXX (XX.X%) | XXX (XX.X%) | | |
| 26 | XXX (XX.X%) | XXX (XX.X%) | | |
| 27 | XXX (XX.X%) | XXX (XX.X%) | | |
| 28 | XXX (XX.X%) | XXX (XX.X%) | | |

Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures. 2. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 13 (FAS) Analysis results of dental examination in the preoperative examination (tooth level) (cont. 1)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Code of LL caries | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 31 | XXX (XX.X%) | XXX (XX.X%) | | |
| 32 | XXX (XX.X%) | XXX (XX.X%) | | |
| 33 | XXX (XX.X%) | XXX (XX.X%) | | |
| 34 | XXX (XX.X%) | XXX (XX.X%) | | |
| 35 | XXX (XX.X%) | XXX (XX.X%) | | |
| 36 | XXX (XX.X%) | XXX (XX.X%) | | |
| 37 | XXX (XX.X%) | XXX (XX.X%) | | |
| 38 | XXX (XX.X%) | XXX (XX.X%) | | |
| Code of LR caries | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 41 | XXX (XX.X%) | XXX (XX.X%) | | |
| 42 | XXX (XX.X%) | XXX (XX.X%) | | |
| 43 | XXX (XX.X%) | XXX (XX.X%) | | |
| 44 | XXX (XX.X%) | XXX (XX.X%) | | |
| 45 | XXX (XX.X%) | XXX (XX.X%) | | |
| 46 | XXX (XX.X%) | XXX (XX.X%) | | |
| 47 | XXX (XX.X%) | XXX (XX.X%) | | |
| 48 | XXX (XX.X%) | XXX (XX.X%) | | |
| Missing (subject level) | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| None | XXX (XX.X%) | XXX (XX.X%) | | |
| With | XXX (XX.X%) | XXX (XX.X%) | | |
| Number of missing (subject l | level) | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 1 | XXX (XX.X%) | XXX (XX.X%) | | |
| 2 | XXX (XX.X%) | XXX (XX.X%) | | |
| | XXX (XX.X%) | XXX (XX.X%) | | |
| Location of missing | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| UR | XXX (XX.X%) | XXX (XX.X%) | | |
| UL | XXX (XX.X%) | XXX (XX.X%) | | |
| LL | XXX (XX.X%) | XXX (XX.X%) | | |
| LR | XXX (XX.X%) | XXX (XX.X%) | | |
| Code of UR missing | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 11 | XXX (XX.X%) | XXX (XX.X%) | | |
| 12 | XXX (XX.X%) | XXX (XX.X%) | | |
| 13 | XXX (XX.X%) | XXX (XX.X%) | | |
| 14 | XXX (XX.X%) | XXX (XX.X%) | | |
| 15 | XXX (XX.X%) | XXX (XX.X%) | | |
| 16 | XXX (XX.X%) | XXX (XX.X%) | | |
| 17 | XXX (XX.X%) | XXX (XX.X%) | | |
| 18 | XXX (XX.X%) | XXX (XX.X%) | | |

Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures.
 Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 13 (FAS) Analysis results of dental examination in the preoperative examination (tooth level) (cont. 2)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Code of UL missing | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 21 | XXX (XX.X%) | XXX (XX.X%) | | |
| 22 | XXX (XX.X%) | XXX (XX.X%) | | |
| 23 | XXX (XX.X%) | XXX (XX.X%) | | |
| 24 | XXX (XX.X%) | XXX (XX.X%) | | |
| 25 | XXX (XX.X%) | XXX (XX.X%) | | |
| 26 | XXX (XX.X%) | XXX (XX.X%) | | |
| 27 | XXX (XX.X%) | XXX (XX.X%) | | |
| 28 | XXX (XX.X%) | XXX (XX.X%) | | |
| Code of LL missing | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 31 | XXX (XX.X%) | XXX (XX.X%) | | |
| 32 | XXX (XX.X%) | XXX (XX.X%) | | |
| 33 | XXX (XX.X%) | XXX (XX.X%) | | |
| 34 | XXX (XX.X%) | XXX (XX.X%) | | |
| 35 | XXX (XX.X%) | XXX (XX.X%) | | |
| 36 | XXX (XX.X%) | XXX (XX.X%) | | |
| 37 | XXX (XX.X%) | XXX (XX.X%) | | |
| 38 | XXX (XX.X%) | XXX (XX.X%) | | |
| Code of LR missing | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 41 | XXX (XX.X%) | XXX (XX.X%) | | |
| 42 | XXX (XX.X%) | XXX (XX.X%) | | |
| 43 | XXX (XX.X%) | XXX (XX.X%) | | |
| 44 | XXX (XX.X%) | XXX (XX.X%) | | |
| 45 | XXX (XX.X%) | XXX (XX.X%) | | |
| 46 | XXX (XX.X%) | XXX (XX.X%) | | |
| 47 | XXX (XX.X%) | XXX (XX.X%) | | |
| 48 | XXX (XX.X%) | XXX (XX.X%) | | |
| Fillings (subject level) | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| None | XXX (XX.X%) | XXX (XX.X%) | | |
| With | XXX (XX.X%) | XXX (XX.X%) | | |
| Number of fillings (subject level) | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 1 | XXX (XX.X%) | XXX (XX.X%) | | |
| 2 | XXX (XX.X%) | XXX (XX.X%) | | |
| | XXX (XX.X%) | XXX (XX.X%) | | |
| Location of filling | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| UR | XXX (XX.X%) | XXX (XX.X%) | | |
| UL | XXX (XX.X%) | XXX (XX.X%) | | |
| LL | XXX (XX.X%) | XXX (XX.X%) | | |
| LR | XXX (XX.X%) | XXX (XX.X%) | | |

1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures.

2. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 13 (FAS) Analysis results of dental examination in the preoperative examination (tooth level) (cont. 3)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Code of UR filling | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 11 | XXX (XX.X%) | XXX (XX.X%) | | |
| 12 | XXX (XX.X%) | XXX (XX.X%) | | |
| 13 | XXX (XX.X%) | XXX (XX.X%) | | |
| 14 | XXX (XX.X%) | XXX (XX.X%) | | |
| 15 | XXX (XX.X%) | XXX (XX.X%) | | |
| 16 | XXX (XX.X%) | XXX (XX.X%) | | |
| 17 | XXX (XX.X%) | XXX (XX.X%) | | |
| 18 | XXX (XX.X%) | XXX (XX.X%) | | |
| Code of UL filling | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 21 | XXX (XX.X%) | XXX (XX.X%) | | |
| 22 | XXX (XX.X%) | XXX (XX.X%) | | |
| 23 | XXX (XX.X%) | XXX (XX.X%) | | |
| 24 | XXX (XX.X%) | XXX (XX.X%) | | |
| 25 | XXX (XX.X%) | XXX (XX.X%) | | |
| 26 | XXX (XX.X%) | XXX (XX.X%) | | |
| 27 | XXX (XX.X%) | XXX (XX.X%) | | |
| 28 | XXX (XX.X%) | XXX (XX.X%) | | |
| Code of LL filling | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 31 | XXX (XX.X%) | XXX (XX.X%) | | |
| 32 | XXX (XX.X%) | XXX (XX.X%) | | |
| 33 | XXX (XX.X%) | XXX (XX.X%) | | |
| 34 | XXX (XX.X%) | XXX (XX.X%) | | |
| 35 | XXX (XX.X%) | XXX (XX.X%) | | |
| 36 | XXX (XX.X%) | XXX (XX.X%) | | |
| 37 | XXX (XX.X%) | XXX (XX.X%) | | |
| 38 | XXX (XX.X%) | XXX (XX.X%) | | |
| Code of LR filling | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 41 | XXX (XX.X%) | XXX (XX.X%) | | |
| 42 | XXX (XX.X%) | XXX (XX.X%) | | |
| 43 | XXX (XX.X%) | XXX (XX.X%) | | |
| 44 | XXX (XX.X%) | XXX (XX.X%) | | |
| 45 | XXX (XX.X%) | XXX (XX.X%) | | |
| 46 | XXX (XX.X%) | XXX (XX.X%) | | |
| 47 | XXX (XX.X%) | XXX (XX.X%) | | |
| 48 | XXX (XX.X%) | XXX (XX.X%) | | |
| Prosthetic teeth or artificial cases (subject level) | rowns | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| None | XXX (XX.X%) | XXX (XX.X%) | | |
| With | XXX (XX.X%) | XXX (XX.X%) | | |

1. Likelihood  $\chi 2$  test or Fisher's exact probability test will be used for group comparison of qualitative measures. 2. Treatment group:  $3M^{TM}$  Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group:  $3M^{TM}$  Filtek<sup>TM</sup> Z350XT.

Table 13 (FAS) Analysis results of dental examination in the preoperative examination (tooth level) (cont. 4)

| Measures | Treatment group | <b>C</b> 1 | Statistics | P value |
|---|---|---|---|---|
| Number of prosthetic teeth or | | | | |
| artificial crowns (subject level) | | | | |
| Cases (Nmiss) | XXX(XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 1 | XXX (XX.X%) | XXX (XX.X%) | | |
| 2 | XXX (XX.X%) | XXX (XX.X%) | | |
| ••• | XXX (XX.X%) | XXX (XX.X%) | | |
| Location of prosthetic tooth or artificial crown | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| UR | XXX (XX.X%) | XXX (XX.X%) | | |
| UL | XXX (XX.X%) | XXX (XX.X%) | | |
| LL | XXX (XX.X%) | XXX (XX.X%) | | |
| LR | XXX (XX.X%) | XXX (XX.X%) | | |
| Code of UR prosthetic tooth or | | | | |
| artificial crown | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 11 | XXX (XX.X%) | XXX (XX.X%) | | |
| 12 | XXX (XX.X%) | XXX (XX.X%) | | |
| 13 | XXX (XX.X%) | XXX (XX.X%) | | |
| 14 | XXX (XX.X%) | XXX (XX.X%) | | |
| 15 | XXX (XX.X%) | XXX (XX.X%) | | |
| 16 | XXX (XX.X%) | XXX (XX.X%) | | |
| 17 | XXX (XX.X%) | XXX (XX.X%) | | |
| 18 | XXX (XX.X%) | XXX (XX.X%) | | |
| Code of UL prosthetic tooth or | | | | |
| artificial crown | | | | |
| Cases (Nmiss) | XXX(XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 21 | XXX (XX.X%) | XXX (XX.X%) | | |
| 22 | XXX (XX.X%) | XXX (XX.X%) | | |
| 23 | XXX (XX.X%) | XXX (XX.X%) | | |
| 24 | XXX (XX.X%) | XXX (XX.X%) | | |
| 25 | XXX (XX.X%) | XXX (XX.X%) | | |
| 26 | XXX (XX.X%) | XXX (XX.X%) | | |
| 27 | XXX (XX.X%) | XXX (XX.X%) | | |
| 28 | XXX (XX.X%) | XXX (XX.X%) | | |
| Code of LL prosthetic tooth or artificial crown | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 31 | XXX (XX.X%) | XXX (XX.X%) | | |
| 32 | XXX (XX.X%) | XXX (XX.X%) | | |
| 33 | XXX (XX.X%) | XXX (XX.X%) | | |
| 34 | XXX (XX.X%) | XXX (XX.X%) | | |
| 35 | XXX (XX.X%) | XXX (XX.X%) | | |
| 36 | XXX (XX.X%) | XXX (XX.X%) | | |
| 37 | XXX (XX.X%) | XXX (XX.X%) | | |
| 38 | XXX (XX.X%) | XXX (XX.X%) | | |
| | (2222270) | (222.22.70) | | |

<sup>2.</sup> Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 13 (FAS) Analysis results of dental examination in the preoperative examination (tooth level) (cont. 5)

| | | •••••••••••••••••••••••••••••••••••••• | | |
|---|---|---|---|---|
| Measures | Treatment group | Control group | Statistics | P value |
| Code of LR prosthetic tooth or | | | | |
| artificial crown | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 41 | XXX (XX.X%) | XXX (XX.X%) | | |
| 42 | XXX (XX.X%) | XXX (XX.X%) | | |
| 43 | XXX (XX.X%) | XXX (XX.X%) | | |
| 44 | XXX (XX.X%) | XXX (XX.X%) | | |
| 45 | XXX (XX.X%) | XXX (XX.X%) | | |
| 46 | XXX (XX.X%) | XXX (XX.X%) | | |
| 47 | XXX (XX.X%) | XXX (XX.X%) | | |
| 48 | XXX (XX.X%) | XXX (XX.X%) | | |

- Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures. 2. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 14 (FAS) Analysis results of pregnancy test in the preoperative examination

| | <b></b> | | | ····· | II |
|---|---|---|---|---|---|
| Measures | Treatment group | Control group | Statistics | P value | |
| Results of pregnancy test | | | | | • |
| Cases (Nmiss) | XXX (XXX) | XXX(XXX) | X.XXXX | X.XXXX | |
| Positive | XXX (XX.X%) | XXX (XX.X%) | | | |
| Negative | XXX (XX.X%) | XXX (XX.X%) | | | |

Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures. 2. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 15 (FAS) Analysis results of oral soft tissue examination in the preoperative examination

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Conduct oral soft tissue examination | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Normality of oral soft tissue | , , | , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Oral soft tissue area | , | , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 1 | XXX (XX.X%) | XXX (XX.X%) | | |
| 2 | XXX (XX.X%) | XXX (XX.X%) | | |
| 2 | XXX (XX.X%) | XXX (XX.X%) | | |
| Examination results area (area level) | 717171 (7171.7170) | 717171 (7171.7170) | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| None | XXX (XX.X%) | XXX (XX.X%) | 21.22222 | 21.21.21.21 |
| 1 | XXX (XX.X%) | XXX(XX.X%) | | |
| 2 | XXX (XX.X%) | XXX(XX.X%) $XXX(XX.X%)$ | | |
| 3 | XXX (XX.X%) | XXX(XX.X%) $XXX(XX.X%)$ | | |
| 4 | | XXX (XX.X%) $XXX (XX.X%)$ | | |
| 5 | XXX (XX.X%)<br>XXX (XX.X%) | | | |
| 6 | XXX (XX.X%) | XXX (XX.X%) | | |
| 7 | ` / | XXX (XX.X%) | | |
| 8 | XXX (XX.X%) | XXX (XX.X%) | | |
| 8<br>9 | XXX (XX.X%) | XXX (XX.X%) | | |
| 10 | XXX (XX.X%) | XXX (XX.X%) | | |
| | XXX (XX.X%) | XXX (XX.X%) | | |
| 11 | XXX (XX.X%) | XXX (XX.X%) | | |
| 12 | XXX (XX.X%) | XXX (XX.X%) | | |
| 13 | XXX (XX.X%) | XXX (XX.X%) | | |
| 14 | XXX (XX.X%) | XXX (XX.X%) | | |
| 15 | XXX (XX.X%) | XXX (XX.X%) | | |
| 16 | XXX (XX.X%) | XXX (XX.X%) | | |
| 17 | XXX (XX.X%) | XXX (XX.X%) | | |
| 18 | XXX (XX.X%) | XXX (XX.X%) | | |
| 19 | XXX (XX.X%) | XXX (XX.X%) | | |
| 20 | XXX (XX.X%) | XXX (XX.X%) | | |
| 21 | XXX (XX.X%) | XXX (XX.X%) | | |
| 22 | XXX (XX.X%) | XXX (XX.X%) | | |
| 23 Dorsum linguae | XXX (XX.X%) | XXX (XX.X%) | | |
| 24 Ventral linguae | XXX (XX.X%) | XXX (XX.X%) | | |
| 25 Apex linguae | XXX (XX.X%) | XXX (XX.X%) | | |
| 26 Lingual margin | XXX (XX.X%) | XXX (XX.X%) | | |
| 27 Tongue base | XXX (XX.X%) | XXX (XX.X%) | | |
| 28 Epiglottis | XXX (XX.X%) | XXX (XX.X%) | | |

- Notes: 1. Likelihood  $\chi$ 2 test or Fisher's exact probability test will be used for group comparison of qualitative measures.
  - 2. Group t-test or Wilcoxon Rank Sum test will be used for group comparison of quantitative measures.
  - 3. For quantitative measures Q1: 25th quantile Q3: 75th quantile.
  - 4. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 15 (FAS) Analysis results of oral soft tissue examination in the preoperative examination (cont.)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Size a (mm) of oral examination | result (area level) | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX. XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Size b (mm) of oral examination | result (area level) | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX. XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Size a*b (mm) of oral examination | on result (area level) | | | |
| XX*XX | XXX (XX.X%) | XXX (XX.X%) | | |
| ••• | XXX (XX.X%) | XXX (XX.X%) | | |
| Clinical significance of oral exar | mination result (area level) | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |

- Notes: 1. Likelihood  $\chi^2$  test or Fisher's exact probability test will be used for group comparison of qualitative measures.
  - 2. Group t-test or Wilcoxon Rank Sum test will be used for group comparison of quantitative measures.
  - 3. For quantitative measures Q1: 25th quantile Q3: 75th quantile.
  - 4. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 16 (FAS) Analysis results of the initial screening in the preoperative examination (tooth level)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Number of teeth passing the | he initial screening criteria (si | abject level) | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 1 | XXX (XX.X%) | XXX (XX.X%) | | |
| 2 | XXX (XX.X%) | XXX (XX.X%) | | |
| 3 | XXX (XX.X%) | XXX (XX.X%) | | |
| 4 | XXX (XX.X%) | XXX (XX.X%) | | |
| 5 | XXX (XX.X%) | XXX (XX.X%) | | |
| Location of diseased tooth | 1 | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| UR | XXX (XX.X%) | XXX (XX.X%) | | |
| UL | XXX (XX.X%) | XXX (XX.X%) | | |
| LL | XXX (XX.X%) | XXX (XX.X%) | | |
| LR | XXX (XX.X%) | XXX (XX.X%) | | |
| Code of UR diseased tootl | h | , , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 11 | XXX (XX.X%) | XXX (XX.X%) | | |
| 12 | XXX (XX.X%) | XXX (XX.X%) | | |
| 13 | XXX (XX.X%) | XXX (XX.X%) | | |
| 14 | XXX (XX.X%) | XXX (XX.X%) | | |
| 15 | XXX (XX.X%) | XXX (XX.X%) | | |
| 16 | XXX (XX.X%) | XXX (XX.X%) | | |
| 17 | XXX (XX.X%) | XXX (XX.X%) | | |
| 18 | XXX (XX.X%) | XXX (XX.X%) | | |
| Code of UL diseased tooth | h | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 21 | XXX (XX.X%) | XXX (XX.X%) | | |
| 22 | XXX (XX.X%) | XXX (XX.X%) | | |
| 23 | XXX (XX.X%) | XXX (XX.X%) | | |
| 24 | XXX (XX.X%) | XXX (XX.X%) | | |
| 25 | XXX (XX.X%) | XXX (XX.X%) | | |
| 26 | XXX (XX.X%) | XXX (XX.X%) | | |
| 27 | XXX (XX.X%) | XXX (XX.X%) | | |
| 28 | XXX (XX.X%) | XXX (XX.X%) | | |

Notes

- 1. Likelihood  $\chi 2$  test or Fisher's exact probability test will be used for group comparison of qualitative measures.
- 2. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 16 (FAS) Analysis results of the initial screening in the preoperative examination (tooth level) (cont.)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Code of LL diseased tooth | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 31 | XXX (XX.X%) | XXX (XX.X%) | | |
| 32 | XXX (XX.X%) | XXX (XX.X%) | | |
| 33 | XXX (XX.X%) | XXX (XX.X%) | | |
| 34 | XXX (XX.X%) | XXX (XX.X%) | | |
| 35 | XXX (XX.X%) | XXX (XX.X%) | | |
| 36 | XXX (XX.X%) | XXX (XX.X%) | | |
| 37 | XXX (XX.X%) | XXX (XX.X%) | | |
| 38 | XXX (XX.X%) | XXX (XX.X%) | | |
| Code of LR diseased tooth | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 41 | XXX (XX.X%) | XXX (XX.X%) | | |
| 42 | XXX (XX.X%) | XXX (XX.X%) | | |
| 43 | XXX (XX.X%) | XXX (XX.X%) | | |
| 44 | XXX (XX.X%) | XXX (XX.X%) | | |
| 45 | XXX (XX.X%) | XXX (XX.X%) | | |
| 46 | XXX (XX.X%) | XXX (XX.X%) | | |
| 47 | XXX (XX.X%) | XXX (XX.X%) | | |
| 48 | XXX (XX.X%) | XXX (XX.X%) | | |

- Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures. 2. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 17 (FAS) Analysis results of cavity preparation of diseased teeth in the screening period

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Location of tooth included in o | cavity preparation | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| UR | XXX (XX.X%) | XXX (XX.X%) | | |
| UL | XXX (XX.X%) | XXX (XX.X%) | | |
| LL | XXX (XX.X%) | XXX (XX.X%) | | |
| LR | XXX (XX.X%) | XXX (XX.X%) | | |
| Code of UR tooth included in | cavity preparation | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 11 | XXX (XX.X%) | XXX (XX.X%) | | |
| 12 | XXX (XX.X%) | XXX (XX.X%) | | |
| 13 | XXX (XX.X%) | XXX (XX.X%) | | |
| 14 | XXX (XX.X%) | XXX (XX.X%) | | |
| 15 | XXX (XX.X%) | XXX (XX.X%) | | |
| 16 | XXX (XX.X%) | XXX (XX.X%) | | |
| 17 | XXX (XX.X%) | XXX (XX.X%) | | |
| 18 | XXX (XX.X%) | XXX (XX.X%) | | |
| Code of UL tooth included in | cavity preparation | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 21 | XXX (XX.X%) | XXX (XX.X%) | | |
| 22 | XXX (XX.X%) | XXX (XX.X%) | | |
| 23 | XXX (XX.X%) | XXX (XX.X%) | | |
| 24 | XXX (XX.X%) | XXX (XX.X%) | | |
| 25 | XXX (XX.X%) | XXX (XX.X%) | | |
| 26 | XXX (XX.X%) | XXX (XX.X%) | | |
| 27 | XXX (XX.X%) | XXX (XX.X%) | | |
| 28 | XXX (XX.X%) | XXX (XX.X%) | | |

<sup>2.</sup> Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 17 (FAS) Analysis results of cavity preparation of diseased teeth in the screening period (cont.)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Code of LL tooth include | d in cavity preparation | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 31 | XXX (XX.X%) | XXX (XX.X%) | | |
| 32 | XXX (XX.X%) | XXX (XX.X%) | | |
| 33 | XXX (XX.X%) | XXX (XX.X%) | | |
| 34 | XXX (XX.X%) | XXX (XX.X%) | | |
| 35 | XXX (XX.X%) | XXX (XX.X%) | | |
| 36 | XXX (XX.X%) | XXX (XX.X%) | | |
| 37 | XXX (XX.X%) | XXX (XX.X%) | | |
| 38 | XXX (XX.X%) | XXX (XX.X%) | | |
| Code of LR tooth include | d in cavity preparation | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 41 | XXX (XX.X%) | XXX (XX.X%) | | |
| 42 | XXX (XX.X%) | XXX (XX.X%) | | X.XXXX |
| 43 | XXX (XX.X%) | XXX (XX.X%) | | |
| 44 | XXX (XX.X%) | XXX (XX.X%) | | |
| 45 | XXX (XX.X%) | XXX (XX.X%) | | |
| 46 | XXX (XX.X%) | XXX (XX.X%) | | |
| 47 | XXX (XX.X%) | XXX (XX.X%) | | |
| 48 | XXX (XX.X%) | XXX (XX.X%) | | |

- Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures. 2. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 18 (FAS) Analysis results of X-ray (periapical radiograph) examination before cavity preparation in the screening period

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| X-ray (periapical radiograph) examina | tion before cavity | | | |
| preparation | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Depth of lesion in X-ray findings | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Shallow dentin | XXX (XX.X%) | XXX (XX.X%) | | |
| Middle dentin | XXX (XX.X%) | XXX (XX.X%) | | |
| Deep dentin | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal or normal X-ray findings | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |

Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures. 2. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 19 (FAS) Analysis results of digital photos before cavity preparation in the screening period

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Take digital photos before cav | vity preparation | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos before cavity | preparation | , , | | |
| Photos of occlusal surface | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos before cavity | preparation | , | | |
| Photos of occlusal surface (wi | | d) | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos before cavity | preparation | , , | | |
| Photos of median occlusion | • | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos before cavity | preparation | | | |
| Photos of antagonist tooth | - | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos before cavity | preparation | | | |
| Photos of buccal surface | • | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos before cavity | preparation | , , | | |
| Photos of lingual surface | • | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos before cavity | | , , | | |
| Other | · • | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |

- Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures. 2. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 20 (FAS) Analysis results of cavity preparation process records in the screening period

| Measures Removed material during the car | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Removed material during the car | vity preparation process | | | |
| Detritus | 7 1 1 | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Removed material during the car | | , | | |
| Original filling | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Removed material during the car | | , | | |
| Thin-wall and low cusps | rity propulation process | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | 71.71.71.71 | 71.7171.717 |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Removed material during the car | , | 7222 (722270) | | |
| Soft scales | vity preparation process | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | 71.71.71.71 | 7.717171 |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Removed material during the car | | AAA(AA.A/0) | | |
| Calculus | vity preparation process | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | Λ.ΛΛΛΛ | Λ.ΛΛΛΛ |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Removed material during the car | · / | $\Lambda\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda/6)$ | | |
| Other | vity preparation process | | | |
| Cases (Nmiss) | VVV (VVV) | VVV (VVV) | X.XXXX | X.XXXX |
| No | XXX (XXX) | XXX (XXX) | Λ.ΛΛΛΛ | Λ.ΛΛΛΛ |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| | XXX (XX.X%) | XXX (XX.X%) | | |
| Local anesthesia applied | VVV (VVV) | VVV (VVV) | v vvvv | vvvvv |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Missing third molar | WWW (WWW) | WWW (WWW) | V VVVV | w www |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Cavity classification | 3/3/3/ (3/3/3/) | 3/3/3/ (3/3/3/) | 37 37373737 | 37 37373737 |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Class I cavities | XXX (XX.X%) | XXX (XX.X%) | | |
| Class II cavities | XXX (XX.X%) | XXX (XX.X%) | | |
| Cavity classification | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| O | XXX (XX.X%) | XXX (XX.X%) | | |
| BO | XXX (XX.X%) | XXX (XX.X%) | | |
| BOL | XXX (XX.X%) | XXX (XX.X%) | | |
| LO | XXX (XX.X%) | XXX (XX.X%) | | |
| MO | XXX (XX.X%) | XXX (XX.X%) | | |
| MOD | XXX (XX.X%) | XXX (XX.X%) | | |
| DO | XXX (XX.X%) | XXX (XX.X%) | | |
| 111011000011000110001100011000110001100011000110001100011000110001100011000110001100011000110001100011000110001 | | | | |

<sup>2.</sup> Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 20 (FAS) Analysis results of cavity preparation process records in the screening period (cont. 1)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Bevel on prepared cavity marg | in | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Bevel angle (degrees) | , | , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean ± SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| O1; O3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Bevel width (mm) | , | , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean ± SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum buccolingual distance | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean ± SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Buccolingual distance betweer | | , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean ± SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Cavity size and maximum buc | | , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean ± SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Cavity size and maximum prox | | | n) | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean ± SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | 1111111111 | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |

Version V1.1

<sup>2.</sup> Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 20 (FAS) Analysis results of cavity preparation process records in the screening period (cont. 2)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Maximum depth after cavity preparation (mm) | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Gingival margin after cavity preparation | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Supragingival | XXX (XX.X%) | XXX (XX.X%) | | |
| Subgingival | XXX (XX.X%) | XXX (XX.X%) | | |
| Not applicable (Class I cavities) | XXX (XX.X%) | XXX (XX.X%) | | |
| Internal line angles of cavity are not rounded en | ough after cavity prep | paration | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Overhang enamel at cavity margin after prepara | ntion | , , , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Cavity bottom | , | , , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Middle and deep dentin | XXX (XX.X%) | XXX (XX.X%) | | |
| (without being close to and not exposing pulp) | , , | , , | | |
| Pulp red or exposed | XXX (XX.X%) | XXX (XX.X%) | | |
| (already or close to be expose pulp) | ` , | ` ' | | |

Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures.
 Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 21 (FAS) Analysis results of digital photos after cavity preparation in the screening period

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Take digital photos after cavity | preparation | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos after cavity pre- | paration | | | |
| Photos of occlusal surface | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos after cavity pre- | paration | | | |
| Photos of occlusal surface (with | h occlusal contacts marked) | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos after cavity pre- | paration | | | |
| Photos of median occlusion | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos after cavity pre- | paration | | | |
| Photos of antagonist tooth | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos after cavity pre- | paration | | | |
| Photos of buccal surface | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos after cavity pre- | paration | , , | | |
| Photos of lingual surface | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos after cavity pre- | | . , | | |
| Other | - | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |

- 1. Likelihood  $\chi 2$  test or Fisher's exact probability test will be used for group comparison of qualitative measures. 2. Treatment group:  $3M^{TM}$  Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group:  $3M^{TM}$  Filtek<sup>TM</sup> Z350XT.

Table 22 (FAS) Analysis results of oral soft tissue examination after cavity preparation in the screening period

| Measures | Treatment group | Control group | | P value |
|---|---|---|---|---|
| Conduct oral soft tissue examination | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Normality of oral soft tissue | , , | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Oral soft tissue area | , | , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 1 | XXX (XX.X%) | XXX (XX.X%) | | |
| 2 | XXX (XX.X%) | XXX (XX.X%) | | |
| _<br> | XXX (XX.X%) | XXX (XX.X%) | | |
| Examination results area (area level) | 11111 (11111170) | 11111 (11111170) | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| None | XXX (XX.X%) | XXX (XX.X%) | | |
| 1 | XXX (XX.X%) | XXX (XX.X%) | | |
| 2 | XXX (XX.X%) | XXX (XX.X%) | | |
| 3 | XXX (XX.X%) | XXX (XX.X%) | | |
| 4 | XXX (XX.X%) | XXX (XX.X%) | | |
| 5 | XXX (XX.X%) | XXX (XX.X%) | | |
| 6 | XXX (XX.X%) | XXX (XX.X%) | | |
| 7 | XXX (XX.X%) | XXX (XX.X%) | | |
| 8 | XXX (XX.X%) | XXX (XX.X%) | | |
| 9 | XXX (XX.X%) | XXX (XX.X%) | | |
| 10 | XXX (XX.X%) | XXX (XX.X%) | | |
| 11 | XXX (XX.X%) | XXX (XX.X%) | | |
| 12 | XXX (XX.X%) | XXX (XX.X%) $XXX (XX.X%)$ | | |
| 13 | XXX (XX.X%) | XXX (XX.X%) $XXX (XX.X%)$ | | |
| 14 | XXX (XX.X%) | XXX (XX.X%) $XXX (XX.X%)$ | | |
| 15 | | | | |
| | XXX (XX.X%) | XXX (XX.X%) | | |
| 16 | XXX (XX.X%) | XXX (XX.X%) | | |
| 17 | XXX (XX.X%) | XXX (XX.X%) | | |
| 18 | XXX (XX.X%) | XXX (XX.X%) | | |
| 19 | XXX (XX.X%) | XXX (XX.X%) | | |
| 20 | XXX (XX.X%) | XXX (XX.X%) | | |
| 21 | XXX (XX.X%) | XXX (XX.X%) | | |
| 22 | XXX (XX.X%) | XXX (XX.X%) | | |
| 23 Dorsum linguae | XXX (XX.X%) | XXX (XX.X%) | | |
| 24 Ventral linguae | XXX (XX.X%) | XXX (XX.X%) | | |
| 25 Apex linguae | XXX (XX.X%) | XXX (XX.X%) | | |
| 26 Lingual margin | XXX (XX.X%) | XXX (XX.X%) | | |
| 27 Tongue base | XXX (XX.X%) | XXX (XX.X%) | | |
| 28 Epiglottis | XXX (XX.X%) | XXX (XX.X%) | | |

- Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures.
  - 2. Group t-test or Wilcoxon Rank Sum test will be used for group comparison of quantitative measures.
  - 3. For quantitative measures Q1: 25th quantile Q3: 75th quantile.
  - 4. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 22 (FAS) Analysis results of oral soft tissue examination after cavity preparation in the screening period (cont.)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Size a (mm) of oral examination | on result (area level) | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean $\pm$ SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Size b (mm) of oral examination | on result (area level) | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean $\pm$ SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Size a*b (mm) of oral examina | ation result (area level) | | | |
| XX*XX | XXX (XX.X%) | XXX (XX.X%) | | |
| ••• | XXX (XX.X%) | XXX (XX.X%) | | |
| Clinical significance of oral ex | camination result (area level | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |

- Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures.
  - 2. Group t-test or Wilcoxon Rank Sum test will be used for group comparison of quantitative measures.
  - 3. For quantitative measures Q1: 25th quantile Q3: 75th quantile.
  - 4. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 23 (FAS) Analysis results of screening results in cavity preparation phase in the screening period (tooth level)

| Passed screening and formally included in the filling phase (subject level) Cases (Nmiss) XXX (XXX) XXX (XXXX) XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | e | P value | Statistics | Control group | Treatment group | Measures |
|---|---|---|---|---|---|---|
| (subject level) Cases (Nmiss) XXX (XXX) XXX (XXXX) XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | Passed screening and formally inclu |
| Cases (Nmiss) XXX (XXX) XXX (XXXX) XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | 81 | |
| No XXX (XX.X%) XXX (XX.X%) Yes XXX (XX.X%) XXX (XX.X%) Location code of formally included tooth: location of diseased tooth XXX (XXX) XXX (XXX) Cases (Nmiss) XXX (XXX.X%) XXX (XX.X%) UL XXX (XX.X%) XXX (XX.X%) LL XXX (XX.X%) XXX (XX.X%) LCoation code of formally included tooth: Code of UR diseased tooth XXX (XXXX) XXX (XXXX) Cases (Nmiss) XXX (XXXX%) XXX (XXXX%) 11 XXX (XX.X%) XXX (XX.X%) 12 XXX (XX.X%) XXX (XX.X%) 13 XXX (XX.X%) XXX (XX.X%) 14 XXX (XX.X%) XXX (XX.X%) 15 XXX (XX.X%) XXX (XX.X%) 16 XXX (XX.X%) XXX (XX.X%) 17 XXX (XX.X%) XXX (XX.X%) 18 XXX (XX.X%) XXX (XX.X%) | XX | X.XXX | X.XXXX | XXX (XXX) | XXX (XXX) | , , |
| Location code of formally included tooth: location of diseased tooth XXX (XXX) XXX (XXX) XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |
| tooth: location of diseased tooth Cases (Nmiss) | | | | XXX (XX.X%) | XXX (XX.X%) | Yes |
| tooth: location of diseased tooth Cases (Nmiss) | | | | | | Location code of formally included |
| UR XXX (XX.X%) XXX (XX.X%) UL XXX (XX.X%) XXX (XX.X%) LL XXX (XX.X%) XXX (XX.X%) LR XXX (XX.X%) XXX (XX.X%) Location code of formally included tooth: Code of UR diseased tooth XXX (XXXX) XXX (XXXX) Cases (Nmiss) XXX (XX.X%) XXX (XX.X%) 11 XXX (XX.X%) XXX (XX.X%) 12 XXX (XX.X%) XXX (XX.X%) 13 XXX (XX.X%) XXX (XX.X%) 14 XXX (XX.X%) XXX (XX.X%) 15 XXX (XX.X%) XXX (XX.X%) 16 XXX (XX.X%) XXX (XX.X%) 17 XXX (XX.X%) XXX (XX.X%) 18 XXX (XX.X%) XXX (XX.X%) | | | | | | |
| UL XXX (XX.X%) XXX (XX.X%) LL XXX (XX.X%) XXX (XX.X%) LR XXX (XX.X%) XXX (XX.X%) Location code of formally included tooth: Code of UR diseased tooth XXX (XXXX) XXX (XXXX) Cases (Nmiss) XXX (XX.X%) XXX (XX.X%) 11 XXX (XX.X%) XXX (XX.X%) 12 XXX (XX.X%) XXX (XX.X%) 13 XXX (XX.X%) XXX (XX.X%) 14 XXX (XX.X%) XXX (XX.X%) 15 XXX (XX.X%) XXX (XX.X%) 16 XXX (XX.X%) XXX (XX.X%) 17 XXX (XX.X%) XXX (XX.X%) 18 XXX (XX.X%) XXX (XX.X%) | ΚX | X.XXX | X.XXXX | XXX (XXX) | XXX (XXX) | Cases (Nmiss) |
| LL XXX (XX.X%) XXX (XX.X%) LR XXX (XX.X%) XXX (XX.X%) Location code of formally included tooth: Code of UR diseased tooth XXX (XXX) XXX (XXXX) Cases (Nmiss) XXX (XX.X%) XXX (XX.X%) 11 XXX (XX.X%) XXX (XX.X%) 12 XXX (XX.X%) XXX (XX.X%) 13 XXX (XX.X%) XXX (XX.X%) 14 XXX (XX.X%) XXX (XX.X%) 15 XXX (XX.X%) XXX (XX.X%) 16 XXX (XX.X%) XXX (XX.X%) 17 XXX (XX.X%) XXX (XX.X%) 18 XXX (XX.X%) XXX (XX.X%) | | | | XXX (XX.X%) | XXX (XX.X%) | UR |
| LR XXX (XX.X%) XXX (XX.X%) Location code of formally included tooth: Code of UR diseased tooth XXX (XXX) XXX (XXXX) Cases (Nmiss) XXX (XX.X%) XXX (XX.X%) 11 XXX (XX.X%) XXX (XX.X%) 12 XXX (XX.X%) XXX (XX.X%) 13 XXX (XX.X%) XXX (XX.X%) 14 XXX (XX.X%) XXX (XX.X%) 15 XXX (XX.X%) XXX (XX.X%) 16 XXX (XX.X%) XXX (XX.X%) 17 XXX (XX.X%) XXX (XX.X%) 18 XXX (XX.X%) XXX (XX.X%) | | | | XXX (XX.X%) | XXX (XX.X%) | UL |
| Location code of formally included tooth: Code of UR diseased tooth XXX (XXX) XXX (XXX) XXX (XXXX) XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | XXX (XX.X%) | XXX (XX.X%) | LL |
| tooth: Code of UR diseased tooth Cases (Nmiss) XXX (XXX) XXX (XXXX) XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | XXX (XX.X%) | XXX (XX.X%) | LR |
| Cases (Nmiss) XXX (XXX) XXX (XXXX) XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |
| 11 XXX (XX.X%) XXX (XX.X%) 12 XXX (XX.X%) XXX (XX.X%) 13 XXX (XX.X%) XXX (XX.X%) 14 XXX (XX.X%) XXX (XX.X%) 15 XXX (XX.X%) XXX (XX.X%) 16 XXX (XX.X%) XXX (XX.X%) 17 XXX (XX.X%) XXX (XX.X%) 18 XXX (XX.X%) XXX (XX.X%) | | | | | | |
| 12 XXX (XX.X%) XXX (XX.X%) 13 XXX (XX.X%) XXX (XX.X%) 14 XXX (XX.X%) XXX (XX.X%) 15 XXX (XX.X%) XXX (XX.X%) 16 XXX (XX.X%) XXX (XX.X%) 17 XXX (XX.X%) XXX (XX.X%) 18 XXX (XX.X%) XXX (XX.X%) | ΚX | X.XXX | X.XXXX | * * | | Cases (Nmiss) |
| 13 XXX (XX.X%) XXX (XX.X%) 14 XXX (XX.X%) XXX (XX.X%) 15 XXX (XX.X%) XXX (XX.X%) 16 XXX (XX.X%) XXX (XX.X%) 17 XXX (XX.X%) XXX (XX.X%) 18 XXX (XX.X%) XXX (XX.X%) | | | | | | |
| 14 XXX (XX.X%) XXX (XX.X%) 15 XXX (XX.X%) XXX (XX.X%) 16 XXX (XX.X%) XXX (XX.X%) 17 XXX (XX.X%) XXX (XX.X%) 18 XXX (XX.X%) XXX (XX.X%) | | | | | | |
| 15 | | | | | | |
| 16 XXX (XX.X%) XXX (XX.X%) 17 XXX (XX.X%) XXX (XX.X%) 18 XXX (XX.X%) XXX (XX.X%) | | | | * | | |
| 17 | | | | | | |
| $18 \qquad \qquad XXX (XX.X\%) \qquad XXX (XX.X\%)$ | | | | | | |
| Location code of formally included | | | | XXX (XX.X%) | XXX (XX.X%) | |
| tooth: Code of UL diseased tooth | | 37 373737 | 37 37373737 | 3/3/3/ (3/3/3/) | 373737 (373737) | |
| Cases (Nmiss) XXX (XXX) XXX (XXX) X.XXXX X.XXXX | ίX | X.XXX | X.XXXX | | | |
| 21 | | | | , | | |
| 22 | | | | | | |
| 23 | | | | | | |
| 24 | | | | | | |
| 25 | | | | | | |
| 26 | | | | , | | |
| | | | | , | | |
| | | | | $\Lambda\Lambda\Lambda$ ( $\Lambda\Lambda.\Lambda$ 70) | $\Lambda\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda\%)$ | |
| Location code of formally included tooth: Code of LL diseased tooth | | | | | | tooth: Code of LL diseased tooth |
| Cases (Nmiss) XXX (XXX) XXX (XXXX X.XXXX X.XXXX | ΚX | X.XXX | X.XXXX | | | |
| $XXX (XX.X\%) \qquad XXX (XX.X\%)$ | | | | | | |
| $XXX (XX.X\%) \qquad XXX (XX.X\%)$ | | | | | | |
| $XXX (XX.X\%) \qquad XXX (XX.X\%)$ | | | | , , | , , | |
| 34 | | | | | | |
| 35 | | | | ` / | ` / | |
| 36 | | | | | | |
| 37 | | | | , | | |
| 38 XXX (XX.X%) XXX (XX.X%) | | | | XXX (XX.X%) | XXX (XX.X%) | 38 |

Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures. 2. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 23 (FAS) Analysis results of screening results in cavity preparation phase in the screening period (tooth level) (cont.)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Location code of forma | ally included tooth: | | | |
| Code of LR diseased to | ooth | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 41 | XXX (XX.X%) | XXX (XX.X%) | | |
| 42 | XXX (XX.X%) | XXX (XX.X%) | | |
| 43 | XXX (XX.X%) | XXX (XX.X%) | | |
| 44 | XXX (XX.X%) | XXX (XX.X%) | | |
| 45 | XXX (XX.X%) | XXX (XX.X%) | | |
| 46 | XXX (XX.X%) | XXX (XX.X%) | | |
| 47 | XXX (XX.X%) | XXX (XX.X%) | | |
| 48 | XXX (XX.X%) | XXX (XX.X%) | | |
| | • / | ` ' | | |

Notes: 1. Likelihood  $\chi^2$  test or Fisher's exact probability test will be used for group comparison of qualitative measures.

<sup>2.</sup> Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 24 (FAS) Analysis results of intraoperative information of all diseased teeth (tooth level)

| Measures | e |
|---|---|
| Cases (Nmiss) XXX (XXX) XXX (XXXX%) XXXX (XXXX%) UR XXX (XXXX%) XXX (XXXX%) XXX (XXXX%) UL XXX (XXXX%) XXX (XXXX%) XXX (XXXX%) LR XXX (XXXX%) XXX (XXXX%) XXX (XXXX%) Information of caries/disease teeth formally included in the study Tooth location code UR XXX (XXXX%) XXX (XXXXX%) Cases (Nmiss) XXX (XXXX%) XXX (XXXX%) XXX (XXXX%) 12 XXX (XXXX%) XXX (XXXX%) 13 XXX (XXXX%) XXX (XXXX%) 14 XXX (XXXX%) XXX (XXXX%) 15 XXX (XXXX%) XXX (XXXX%) 16 XXX (XXXX%) XXX (XXXX%) 17 XXX (XXXX%) XXX (XXXX%) 18 XXX (XXXX%) XXX (XXXX%) 19 XXX (XXXXX%) XXX (XXXXX%) 10 XXX (XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| UR | XX |
| UL XXX (XX.X%) XXX (XX.X%) LL XXX (XX.X%) XXX (XX.X%) LR XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study XXX (XXX) XXX (XXXX) Cases (Nmiss) XXX (XXX.X%) XXX (XX.X%) 11 XXX (XX.X%) XXX (XX.X%) 12 XXX (XX.X%) XXX (XX.X%) 13 XXX (XX.X%) XXX (XX.X%) 14 XXX (XX.X%) XXX (XX.X%) 15 XXX (XX.X%) XXX (XX.X%) 16 XXX (XX.X%) XXX (XX.X%) 17 XXX (XX.X%) XXX (XX.X%) 18 XXX (XX.X%) XXX (XX.X%) 10 XXX (XX.X%) XXX (XX.X%) 11 XXX (XX.X%) XXX (XX.X%) 12 XXX (XX.X%) XXX (XX.X%) 13 XXX (XX.X%) XXX (XX.X%) 14 XXX (XX.X%) XXX (XX.X%) 15 XXX (XX.X%) XXX (XX.X%) 16 XXX (XX.X%) XXX (XX.X%) 17 | |
| LL XXX (XX.X%) XXX (XX.X%) LR XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code UR Cases (Nmiss) XXX (XXXX) XXX (XXXX%) 11 XXX (XX.X%) XXX (XX.X%) 12 XXX (XX.X%) XXX (XX.X%) 13 XXX (XX.X%) XXX (XX.X%) 14 XXX (XX.X%) XXX (XX.X%) 15 XXX (XX.X%) XXX (XX.X%) 16 XXX (XX.X%) XXX (XX.X%) 17 XXX (XX.X%) XXX (XX.X%) 18 XXX (XX.X%) XXX (XX.X%) 19 XXX (XX.X%) XXX (XX.X%) 10 XXX (XX.X%) XXX (XX.X%) 11 XXX (XX.X%) XXX (XX.X%) 12 XXX (XX.X%) XXX (XX.X%) 13 XXX (XX.X%) XXX (XX.X%) 14 XXX (XX.X%) XXX (XX.X%) 15 XXX (XX.X%) XXX (XX.X%) 16 XXX (XX.X%) XXX (XX.X%) 17 XXX (XX | |
| LR XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code UR Cases (Nmiss) XXX (XXX) XXX (XXXX%) 11 XXX (XX.X%) XXX (XX.X%) 12 XXX (XX.X%) XXX (XX.X%) 13 XXX (XX.X%) XXX (XX.X%) 14 XXX (XX.X%) XXX (XX.X%) 15 XXX (XX.X%) XXX (XX.X%) 16 XXX (XX.X%) XXX (XX.X%) 17 XXX (XX.X%) XXX (XX.X%) 18 XXX (XX.X%) XXX (XX.X%) 18 XXX (XX.X%) XXX (XX.X%) 10 XXX (XX.X%) XXX (XX.X%) 11 XXX (XX.X%) XXX (XX.X%) 12 XXX (XX.X%) XXX (XX.X%) 13 XXX (XX.X%) XXX (XX.X%) 14 XXX (XX.X%) XXX (XX.X%) 15 XXX (XX.X%) XXX (XX.X%) 16 XXX (XX.X%) XXX (XX.X%) 17 XXX (XX.X%) XXX (XX.XX 21 | |
| Information of caries/disease teeth formally included in the study Tooth location code UR Cases (Nmiss) | |
| Tooth location code UR Cases (Nmiss) XXX (XXX) XXX (XXXX%) XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| Cases (Nmiss) XXX (XXX) XXX (XXXX) XXXX XXXX 11 XXX (XXXX%) XXX (XXXX%) XXX (XXXX%) 12 XXX (XXXX%) XXX (XXXX%) XXX (XXXX%) 13 XXX (XXXX%) XXX (XXXX%) XXX (XXXX%) 14 XXX (XXXX%) XXX (XXXX%) XXX (XXXX%) 15 XXX (XXXX%) XXX (XXXX%) XXX (XXXX%) 16 XXX (XXXX%) XXX (XXXX%) XXX (XXXX%) 18 XXX (XXXX%) XXX (XXXX%) XXX (XXXXX 19 XXX (XXXXX XXX (XXXXXX XXX (XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| 11 XXX (XX.X%) XXX (XX.X%) 12 XXX (XX.X%) XXX (XX.X%) 13 XXX (XX.X%) XXX (XX.X%) 14 XXX (XX.X%) XXX (XX.X%) 15 XXX (XX.X%) XXX (XX.X%) 16 XXX (XX.X%) XXX (XX.X%) 17 XXX (XX.X%) XXX (XX.X%) 18 XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code UL XXX (XX.X%) XXX (XX.X%) 21 XXX (XX.X%) XXX (XX.X%) 22 XXX (XX.X%) XXX (XX.X%) 23 XXX (XX.X%) XXX (XX.X%) 24 XXX (XX.X%) XXX (XX.X%) 25 XXX (XX.X%) XXX (XX.X%) 26 XXX (XX.X%) XXX (XX.X%) 27 XXX (XX.X%) XXX (XX.X%) 28 XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code LL | XX |
| 12 XXX (XX.X%) XXX (XX.X%) 13 XXX (XX.X%) XXX (XX.X%) 14 XXX (XX.X%) XXX (XX.X%) 15 XXX (XX.X%) XXX (XX.X%) 16 XXX (XX.X%) XXX (XX.X%) 17 XXX (XX.X%) XXX (XX.X%) 18 XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code UL XXX (XX.X%) XXX (XX.X%) 21 XXX (XX.X%) XXX (XX.X%) 22 XXX (XX.X%) XXX (XX.X%) 23 XXX (XX.X%) XXX (XX.X%) 24 XXX (XX.X%) XXX (XX.X%) 25 XXX (XX.X%) XXX (XX.X%) 26 XXX (XX.X%) XXX (XX.X%) 27 XXX (XX.X%) XXX (XX.X%) 28 XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code LL | |
| 13 XXX (XX.X%) XXX (XX.X%) 14 XXX (XX.X%) XXX (XX.X%) 15 XXX (XX.X%) XXX (XX.X%) 16 XXX (XX.X%) XXX (XX.X%) 17 XXX (XX.X%) XXX (XX.X%) 18 XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code UL XXX (XXXX) XXX (XXXXX) 21 XXX (XXXX%) XXX (XXXX%) 22 XXX (XXXX%) XXX (XXXX%) 23 XXX (XXXX%) XXX (XXXX%) 24 XXX (XXXX%) XXX (XXXX%) 25 XXX (XXXX%) XXX (XXXX%) 26 XXX (XXXX%) XXX (XXXX%) 27 XXX (XXXX%) XXX (XXXX%) 28 XXX (XXXX%) XXX (XXXX%) Information of caries/disease teeth formally included in the study Tooth location code LL | |
| 14 XXX (XX.X%) XXX (XX.X%) 15 XXX (XX.X%) XXX (XX.X%) 16 XXX (XX.X%) XXX (XX.X%) 17 XXX (XX.X%) XXX (XX.X%) 18 XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code UL XXX (XXXX) XXX (XXXXX) 21 XXX (XX.X%) XXX (XX.X%) 22 XXX (XX.X%) XXX (XX.X%) 23 XXX (XX.X%) XXX (XX.X%) 24 XXX (XX.X%) XXX (XX.X%) 25 XXX (XX.X%) XXX (XX.X%) 26 XXX (XX.X%) XXX (XX.X%) 27 XXX (XX.X%) XXX (XX.X%) 28 XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code LL | |
| 15 XXX (XX.X%) XXX (XX.X%) 16 XXX (XX.X%) XXX (XX.X%) 17 XXX (XX.X%) XXX (XX.X%) 18 XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code UL Cases (Nmiss) XXX (XXXX) XXX (XXXX%) 21 XXX (XX.X%) XXX (XX.X%) 22 XXX (XXXX%) XXX (XXXX%) 23 XXX (XXXX%) XXX (XXXX%) 24 XXX (XXXX%) XXX (XXXX%) 25 XXX (XXXX%) XXX (XXXX%) 26 XXX (XXXX%) XXX (XXXX%) 27 XXX (XXXX%) XXX (XXXX%) 28 XXX (XXXXX%) XXX (XXXXX%) Information of caries/disease teeth formally included in the study Tooth location code LL | |
| 16 XXX (XX.X%) XXX (XX.X%) 17 XXX (XX.X%) XXX (XX.X%) 18 XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code UL Cases (Nmiss) XXX (XXXX) XXX (XXXXX) 21 XXX (XX.X%) XXX (XX.X%) 22 XXX (XXXX%) XXX (XXXX%) 23 XXX (XXXX%) XXX (XXXX%) 24 XXX (XXXX%) XXX (XXXX%) 25 XXX (XXXX%) XXX (XXXX%) 26 XXX (XXXX%) XXX (XXXX%) 27 XXX (XXXX%) XXX (XXXX%) 28 XXX (XXXX%) XXX (XXXX%) Information of caries/disease teeth formally included in the study Tooth location code LL XXX (XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| 17 XXX (XX.X%) XXX (XX.X%) 18 XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code UL Cases (Nmiss) XXX (XXXX) XXX (XXXXX) 21 XXX (XX.X%) XXX (XX.X%) 22 XXX (XX.X%) XXX (XX.X%) 23 XXX (XX.X%) XXX (XX.X%) 24 XXX (XX.X%) XXX (XX.X%) 25 XXX (XX.X%) XXX (XX.X%) 26 XXX (XX.X%) XXX (XX.X%) 27 XXX (XX.X%) XXX (XX.X%) 28 XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code LL | |
| 18 XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code UL Cases (Nmiss) XXX (XXX) XXX (XXXX%) XXX (XXXXX%) 21 XXX (XXXX%) XXX (XXXX%) XXX (XXXXX%) 22 XXX (XXXXX%) XXX (XXXXX%) XXX (XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| Information of caries/disease teeth formally included in the study Tooth location code UL Cases (Nmiss) XXX (XXX) XXX (XXX) X.XXX X.XX 21 XXX (XX.X%) XXX (XX.X%) 22 XXX (XX.X%) XXX (XX.X%) 23 XXX (XX.X%) XXX (XX.X%) 24 XXX (XX.X%) XXX (XX.X%) 25 XXX (XX.X%) XXX (XX.X%) 26 XXX (XX.X%) XXX (XX.X%) 27 XXX (XX.X%) XXX (XX.X%) 28 XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code LL | |
| Tooth location code UL Cases (Nmiss) XXX (XXX) XXX (XXXX) X.XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| 21 XXX (XX.X%) XXX (XX.X%) 22 XXX (XX.X%) XXX (XX.X%) 23 XXX (XX.X%) XXX (XX.X%) 24 XXX (XX.X%) XXX (XX.X%) 25 XXX (XX.X%) XXX (XX.X%) 26 XXX (XX.X%) XXX (XX.X%) 27 XXX (XX.X%) XXX (XX.X%) 28 XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code LL | |
| 22 XXX (XX.X%) XXX (XX.X%) 23 XXX (XX.X%) XXX (XX.X%) 24 XXX (XX.X%) XXX (XX.X%) 25 XXX (XX.X%) XXX (XX.X%) 26 XXX (XX.X%) XXX (XX.X%) 27 XXX (XX.X%) XXX (XX.X%) 28 XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code LL | XX |
| 23 XXX (XX.X%) XXX (XX.X%) 24 XXX (XX.X%) XXX (XX.X%) 25 XXX (XX.X%) XXX (XX.X%) 26 XXX (XX.X%) XXX (XX.X%) 27 XXX (XX.X%) XXX (XX.X%) 28 XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code LL | |
| 24 XXX (XX.X%) XXX (XX.X%) 25 XXX (XX.X%) XXX (XX.X%) 26 XXX (XX.X%) XXX (XX.X%) 27 XXX (XX.X%) XXX (XX.X%) 28 XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code LL | |
| 25 XXX (XX.X%) XXX (XX.X%) 26 XXX (XX.X%) XXX (XX.X%) 27 XXX (XX.X%) XXX (XX.X%) 28 XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code LL | |
| 26 XXX (XX.X%) XXX (XX.X%) 27 XXX (XX.X%) XXX (XX.X%) 28 XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code LL | |
| 27 XXX (XX.X%) XXX (XX.X%) 28 XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code LL | |
| 28 XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code LL | |
| 28 XXX (XX.X%) XXX (XX.X%) Information of caries/disease teeth formally included in the study Tooth location code LL | |
| Tooth location code LL | |
| Cases (Nmiss) XXX (XXX) XXX (XXX) X.XXX X.XX | |
| | XX |
| $XXX (XX.X\%) \qquad XXX (XX.X\%)$ | |
| XXX (XX.X%) XXX (XX.X%) | |
| $XXX (XX.X\%) \qquad XXX (XX.X\%)$ | |
| $XXX (XX.X\%) \qquad XXX (XX.X\%)$ | |
| 35 XXX (XX.X%) XXX (XX.X%) | |
| 36 XXX (XX.X%) XXX (XX.X%) | |
| 37 XXX (XX.X%) XXX (XX.X%) | |
| 38 | |
| Information of caries/disease teeth formally included in the study Tooth location code LR | |
| Cases (Nmiss) XXX (XXX) XXX (XXX) X.XXXX X.XX | XX |
| 41 $XXX (XX.X\%)$ $XXX (XX.X\%)$ | 1/1 |
| 44 | |
| 45 | |
| 46 | |
| 47 | |
| 48 XXX (XX.X%) XXX (XX.X%) | |

Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures. 2. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 24 (FAS) Analysis results of intraoperative information of all diseased teeth (tooth level) (cont.)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Other disease teeth that not inc | cluded are treated at the s | ame time | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Location of caries/disease teet | h passing inclusion/exclu | usion criteria but not inclu | ıded | |
| in the study name of product to | o be used | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 3M <sup>TM</sup> Filtek <sup>TM</sup> Z350XT | XXX (XX.X%) | XXX (XX.X%) | | |
| Other | XXX (XX.X%) | XXX (XX.X%) | | |
| Not restored | XXX (XX.X%) | XXX (XX.X%) | | |

Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures.

<sup>2.</sup> Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 25 (FAS) Analysis results of intraoperative records

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| The name of product to be used is | s Filtek <sup>TM</sup> Bulk Fill Poste | erior Restorative | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Name of product to be used: Filte | kTM Z350XT | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Code of investigational device to | | , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| XXX | XXX (XX.X%) | XXX (XX.X%) | | |
| | XXX (XX.X%) | XXX (XX.X%) | | |
| Shade selections for the treatment | t group in the study | ` , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| A1 | XXX (XX.X%) | XXX (XX.X%) | | |
| A2 | XXX (XX.X%) | XXX (XX.X%) | | |
| A3 | XXX (XX.X%) | XXX (XX.X%) | | |
| B1 | XXX (XX.X%) | XXX (XX.X%) | | |
| C2 | XXX (XX.X%) | XXX (XX.X%) | | |
| Shade selections for the control g | , , | , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| A1B | XXX (XX.X%) | XXX (XX.X%) | | |
| A2B | XXX (XX.X%) | XXX (XX.X%) | | |
| A3B | XXX (XX.X%) | XXX (XX.X%) | | |
| A3.5B | XXX (XX.X%) | XXX (XX.X%) | | |
| B1B | XXX (XX.X%) | XXX (XX.X%) | | |
| C2B | XXX (XX.X%) | XXX (XX.X%) | | |
| Filling time (min) | , | , , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean $\pm$ SD | | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Cover pulp or base | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Rubber dam used | . , | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |

- Notes: 1. Likelihood  $\chi^2$  test or Fisher's exact probability test will be used for group comparison of qualitative measures.
  - 2. Group t-test or Wilcoxon Rank Sum test will be used for group comparison of quantitative measures.
  - 3. For quantitative measures Q1: 25th quantile Q3: 75th quantile.
  - 4. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.
  - 5. Filling time = ending time of filling starting time of filling.

Table 25 (FAS) Analysis results of intraoperative records (cont. 1)

| | Table 25 (1715) Analysis results of metaoperative records (cont. 1) | | | |
|---|---|---|---|---|
| Measures | Treatment group | Control group | Statistics | P value |
| Matrix band placed | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Not applicable | XXX (XX.X%) | XXX (XX.X%) | | |
| Brand of adhesive system | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 3M ESPE Single Bond | XXX (XX.X%) | XXX (XX.X%) | | |
| Universal Adhesive | | | | |
| Other | XXX (XX.X%) | XXX (XX.X%) | | |
| Curing time of adhesive | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 10 s | XXX (XX.X%) | XXX (XX.X%) | | |
| Other (seconds) | XXX (XX.X%) | XXX (XX.X%) | | |
| Number of resin layers | | | | |
| Cases (Nmiss) | XXX(XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 1 | XXX (XX.X%) | XXX (XX.X%) | | |
| 2 | XXX (XX.X%) | XXX (XX.X%) | | |
| 3 | XXX (XX.X%) | XXX (XX.X%) | | |
| 4 | XXX (XX.X%) | XXX (XX.X%) | | |
| 5 | XXX (XX.X%) | XXX (XX.X%) | | |
| Thickness of 1st layer (mm) | | | | |
| Cases (Nmiss) | XXX(XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Thickness of 2nd layer (mm) | | | | |
| Cases (Nmiss) | XXX(XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Thickness of 3rd layer (mm) | | | | |
| Cases (Nmiss) | XXX(XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Thickness of 4th layer (mm) | | | | |
| Cases (Nmiss) | XXX(XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |

Notes:

- 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures.
- 2. Group t-test or Wilcoxon Rank Sum test will be used for group comparison of quantitative measures.
- 3. For quantitative measures Q1: 25th quantile Q3: 75th quantile.
- $\text{4. Treatment group: } 3M^{\text{TM}} \text{ Filtek}^{\text{TM}} \text{ Bulk Fill Posterior Restorative; Control group: } 3M^{\text{TM}} \text{ Filtek}^{\text{TM}} \text{ Z350XT.}$

Table 25 (FAS) Analysis results of intraoperative records (cont. 2)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Thickness of 5th layer (mm) | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | x xxxx | X.XXXX |
| Mean ± SD | $XX.XX \pm XX.XX$ | | | Λ.Α.Α.Α.Α. |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | | | |
| Minimum; Maximum | XX.XX; XX.XX | | | |
| Curing method | 727.771, 727.771 | 71717171, 71717171 | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Light Cure | XXX (XX.X%) | XXX (XX.X%) | 11.11111111 | 71.72.1717 |
| Other | XXX (XX.X%) | XXX (XX.X%) | | |
| Brand of curing light | 712121 (7121.2170) | 71.71 (71.71.70) | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 3Mtm Elipar S10 LED Curing Light | XXX (XX.X%) | XXX (XX.X%) | 71.71717171 | 21.21.21.21 |
| Other | XXX (XX.X%) | XXX (XX.X%) | | |
| Output power of curing light measured before | 70.27 (70.71.70) | 71.71 (71.71.70) | | |
| each curing (Mw/cm <sup>2</sup> ) | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean ± SD | $XX.XX \pm XX.XX$ | , , | | Λ.Α.Α.Α.Α.Α. |
| Median | XX.XX ± XX.XX<br>XX.XX | XX.XX ± XX.XZ<br>XX.XX | Y. | |
| Q1; Q3 | XX.XX; XX.XX | | | |
| Minimum; Maximum | XX.XX; XX.XX | | | |
| Cavity type of diseased tooth | $\Lambda\Lambda.\Lambda\Lambda$ , $\Lambda\Lambda.\Lambda\Lambda$ | $\Lambda\Lambda.\Lambda\Lambda$ , $\Lambda\Lambda.\Lambda\Lambda$ | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Class I cavities | XXX (XXX) | XXX (XX.X%) | Α.ΑΑΑΑ | Λ.Α.Α.Α.Α.Α. |
| Class II cavities | XXX (XX.X%) | XXX (XX.X%) | | |
| Curing time of 1st resin layer - Class I cavities | MM(MM.M70) | AAA (AA.A70) | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 20 s | XXX (XX.X%) | XXX (XX.X%) | Α.ΑΑΑΑ | Λ.Α.Α.Α.Α.Α. |
| Other (seconds) | XXX (XX.X%)<br>XXX (XX.X%) | XXX (XX.X%) | | |
| Curing time of 1st resin layer | $\Lambda\Lambda\Lambda$ ( $\Lambda\Lambda.\Lambda$ /0) | $\Lambda\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda/0)$ | | |
| Other (seconds) - Class I cavities | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean ± SD | $XX.XX \pm XX.XX$ | | | Λ.ΛΛΛΛ |
| Median | XX.XX ± XX.XX | XX.XX ± XX.XX | ı | |
| Q1; Q3 | XX.XX; XX.XX | | | |
| Minimum; Maximum | XX.XX; XX.XX | | | |
| Curing time of 2nd resin layer - Class I cavities | | $\Lambda\Lambda.\Lambda\Lambda$ , $\Lambda\Lambda.\Lambda\Lambda$ | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 20 s | XXX (XXX)<br>XXX (XX.X%) | XXX (XX.X%) | Λ.ΛΛΛΛ | Λ.ΛΛΛΛ |
| Other (seconds) | XXX (XX.X%) $XXX (XX.X%)$ | XXX (XX.X%) | | |
| Curing time of 2nd resin layer | $\Lambda\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda/0)$ | $\Lambda\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda/0)$ | | |
| Other (seconds) - Class I cavities | | | | |
| Cases (Nmiss) | XXX (XXX) | VVV (VVV) | vvvvv | X.XXXX |
| Mean ± SD | ` / | XXX (XXX) | X.XXXX | Λ.ΛΛΛΛ |
| | $XX.XX \pm XX.XX$ | | 7 | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |

<sup>2.</sup> Group t-test or Wilcoxon Rank Sum test will be used for group comparison of quantitative measures.

<sup>3.</sup> For quantitative measures Q1: 25th quantile Q3: 75th quantile.

<sup>4.</sup> Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 25 (FAS) Analysis results of intraoperative records (cont. 3)

| | •••• | | | |
|---|---|---|---|---|
| Measures | Treatment group | | | |
| Curing time of 1st layer on occlusal surface - | | | | |
| Class II cavities | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 10 s | XXX (XX.X%) | | | |
| Other (seconds) | XXX (XX.X%) | XXX (XX.X%) | | |
| Curing time of 1st layer on occlusal surface | , | , | | |
| Other (seconds) - Class II cavities | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean $\pm$ SD | | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | | | |
| Curing time of 1st layer on buccal surface - | · | • | | |
| Class II cavities | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 10 s | XXX (XX.X%) | | | |
| Other (seconds) | XXX (XX.X%) | XXX (XX.X%) | | |
| Curing time of 1st layer on buccal surface | | | | |
| Other (seconds) - Class II cavities | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Curing time of 1st layer on lingual surface - | | | | |
| Class II cavities | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 10 s | XXX (XX.X%) | XXX (XX.X%) | | |
| Other (seconds) | XXX (XX.X%) | XXX (XX.X%) | | |
| Curing time of 1st layer on lingual surface | | | | |
| Other (seconds) - Class II cavities | | | | |
| Cases (Nmiss) | XXX(XXX) | \ / | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Curing time of 2nd layer on occlusal surface - | | | | |
| Class II cavities | | | | |
| Cases (Nmiss) | XXX(XXX) | | X.XXXX | X.XXXX |
| 10 s | XXX (XX.X%) | XXX (XX.X%) | | |
| Other (seconds) | XXX (XX.X%) | XXX (XX.X%) | | |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |
| Curing time of 2nd layer on occlusal surface | | | | |
| Other (seconds) - Class II cavities | | | | |
| Cases (Nmiss) | XXX(XXX) | , , | X.XXXX | X.XXXX |
| $Mean \pm SD$ | | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |

- Notes: 1. Likelihood  $\chi^2$  test or Fisher's exact probability test will be used for group comparison of qualitative measures.
  - 2. Group t-test or Wilcoxon Rank Sum test will be used for group comparison of quantitative measures.
  - 3. For quantitative measures Q1: 25th quantile Q3: 75th quantile.
  - 4. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 25 (FAS) Analysis results of intraoperative records (cont. 4)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Curing time of 2nd layer on bu | accal surface - Class II cavities | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 10 s | XXX (XX.X%) | XXX (XX.X%) | | |
| Other (seconds) | XXX (XX.X%) | XXX (XX.X%) | | |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |
| Curing time of 2nd layer on bu | | , | | |
| Other (seconds) - Class II cavi | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean ± SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| | ngual surface - Class II cavities | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 10 s | XXX (XX.X%) | XXX (XX.X%) | | |
| Other (seconds) | XXX (XX.X%) | XXX (XX.X%) | | |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |
| Curing time of 2nd layer on lin | | 71711 (7171.7170) | | |
| Other (seconds) - Class II cavi | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean ± SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | 71.7171717 | 21.22222 |
| Median | XX.XX = XX.XX<br>XX.XX | XX.XX ± XX.XX<br>XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Curing time of 1st layer - Clas | - | MMM, MMM | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 20 s | XXX(XXX) $XXX(XX.X%)$ | XXX (XXX)<br>XXX (XX.X%) | Α.ΑΑΑΑ | Λ.ΛΛΛΛ |
| | XXX (XX.X%) $XXX (XX.X%)$ | XXX (XX.X%) $XXX (XX.X%)$ | | |
| Other (seconds) Curing time of 1st layer | $\Lambda\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda/0)$ | $\Lambda\Lambda\Lambda$ ( $\Lambda\Lambda.\Lambda$ /0) | | |
| | tina | | | |
| Other (seconds) - Class II cavi | | VVV (VVV) | vvvvv | v vvvv |
| Cases (Nmiss)<br>Mean ± SD | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Curing time of 2nd layer - Cla | | VVV (VVVV) | 37.37373737 | 37.37373737 |
| Cases (Nmiss) | | XXX (XXX) | X.XXXX | X.XXXX |
| 20 s | XXX (XX.X%) | XXX (XX.X%) | | |
| Other (seconds) | XXX (XX.X%) | XXX (XX.X%) | | |
| Curing time of 2nd layer | | | | |
| Other (seconds) - Class II cavi | | ****************************** | ** ****** | ** ***** |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean $\pm$ SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |

- Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures.
  - 2. Group t-test or Wilcoxon Rank Sum test will be used for group comparison of quantitative measures.
  - 3. For quantitative measures Q1: 25th quantile Q3: 75th quantile.
  - 4. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 25 (FAS) Analysis results of intraoperative records (cont. 5)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Curing time of 3rd layer - Class I | II cavities | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 20 s | XXX (XX.X%) | XXX (XX.X%) | | |
| Other (seconds) | XXX (XX.X%) | XXX (XX.X%) | | |
| Curing time of 3rd layer | , | , | | |
| Other (seconds) - Class II cavitie | es | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean ± SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| * ' * | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Curing time of 4th layer - Class I | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 20 s | XXX (XX.X%) | XXX (XX.X%) | | |
| Other (seconds) | XXX (XX.X%) | XXX (XX.X%) | | |
| Curing time of 4th layer | ( | () | | |
| Other (seconds) - Class II cavitie | es. | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean $\pm$ SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | 120121212 | 1111111111 |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Curing time of 5th layer - Class I | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 20 s | XXX (XX.X%) | XXX (XX.X%) | | |
| Other (seconds) | XXX (XX.X%) | XXX (XX.X%) | | |
| Curing time of 5th layer | , | , | | |
| Other (seconds) - Class II cavitie | es | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean $\pm$ SD | $XX.XX \pm XX.XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Occlusion adjustment after filling | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Occlusal contact | XXX (XX.X%) | XXX (XX.X%) | | |
| No occlusal contact | XXX (XX.X%) | XXX (XX.X%) | | |
| Cusps of antagonist tooth pressir | , | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Brand of Polishing System to be | | 11111 (11111179) | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 3M <sup>TM</sup> Sof-lex Finishing and<br>Polishing System | | XXX (XX.X%) | | |
| Other | XXX (XX.X%) | XXX (XX.X%) | | |

- Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures.
  - 2. Group t-test or Wilcoxon Rank Sum test will be used for group comparison of quantitative measures.
  - 3. For quantitative measures Q1: 25th quantile Q3: 75th quantile.
  - 4. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 26 (FAS) Analysis results of digital photos taken immediately after the filling procedure

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Take digital photos immediately | after filling | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos | , , | , | | |
| Photos of occlusal surface | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos | | , , | | |
| Photos of occlusal surface (with | occlusal contacts marked) | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos | , | , | | |
| Photos of median occlusion | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos | , | , | | |
| Photos of antagonist tooth | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos | , , | , , | | |
| Photos of buccal surface | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos | , | , | | |
| Photos of lingual surface | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos | , | , | | |
| Other | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |

Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures. 2. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 27 (FAS) Analysis results of oral soft tissue examination in the filling procedure

| Measures | | Control group | | |
|---|---|---|---|---|
| Conduct oral soft tissue exam | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Normality of oral soft tissue | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Oral soft tissue area | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 1 | XXX (XX.X%) | | | |
| 2 | XXX (XX.X%) | · | | |
| | XXX (XX.X%) | XXX (XX.X%) | | |
| Examination results area (area | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| None | XXX (XX.X%) | XXX (XX.X%) | | |
| 1 | XXX (XX.X%) | XXX (XX.X%) | | |
| 2 | XXX (XX.X%) | XXX (XX.X%) | | |
| 3 | XXX (XX.X%) | XXX (XX.X%) | | |
| 4 | XXX (XX.X%) | XXX (XX.X%) | | |
| 5 | XXX (XX.X%) | XXX (XX.X%) | | |
| 6 | XXX (XX.X%) | XXX (XX.X%) | | |
| 7 | XXX (XX.X%) | XXX (XX.X%) | | |
| 8 | XXX (XX.X%) | XXX (XX.X%) | | |
| 9 | XXX (XX.X%) | XXX (XX.X%) | | |
| 10 | XXX (XX.X%) | XXX (XX.X%) | | |
| 11 | XXX (XX.X%) | XXX (XX.X%) | | |
| 12 | XXX (XX.X%) | XXX (XX.X%) | | |
| 13 | XXX (XX.X%) | XXX (XX.X%) | | |
| 14 | XXX (XX.X%) | XXX (XX.X%) | | |
| 15 | XXX (XX.X%) | XXX (XX.X%) | | |
| 16 | XXX (XX.X%) | XXX (XX.X%) | | |
| 17 | XXX (XX.X%) | XXX (XX.X%) | | |
| 18 | XXX (XX.X%) | XXX (XX.X%) | | |
| 19 | XXX (XX.X%) | XXX (XX.X%) | | |
| 20 | XXX (XX.X%) | XXX (XX.X%) | | |
| 21 | XXX (XX.X%) | XXX (XX.X%) | | |
| 22 | XXX (XX.X%) | XXX (XX.X%) | | |
| 23 Dorsum linguae | XXX (XX.X%) | XXX (XX.X%) | | |
| 24 Ventral linguae | XXX (XX.X%) | XXX (XX.X%) | | |
| 25 Apex linguae | XXX (XX.X%) | XXX (XX.X%) | | |
| 26 Lingual margin | XXX (XX.X%) | XXX (XX.X%) | | |
| 27 Tongue base | XXX (XX.X%) | XXX (XX.X%) | | |
| 28 Epiglottis | XXX (XX.X%) | XXX (XX.X%) | | |

<sup>2.</sup> Group t-test or Wilcoxon Rank Sum test will be used for group comparison of quantitative measures.

<sup>3.</sup> For quantitative measures Q1: 25th quantile Q3: 75th quantile.

<sup>4.</sup> Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 27 (FAS) Analysis results of oral soft tissue examination during the filling procedure (cont.)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Size a (mm) of oral examination | on result (area level) | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean $\pm$ SD | $XX.XX \pm XX. XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Size b (mm) of oral examination | on result (area level) | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean $\pm$ SD | $XX.XX \pm XX. XX$ | $XX.XX \pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Size a*b (mm) of oral examina | ation result (area level) | | | |
| XX*XX | XXX (XX.X%) | XXX (XX.X%) | | |
| ••• | XXX (XX.X%) | XXX (XX.X%) | | |
| Clinical significance of oral ex | camination result (area level) | ) | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |

- Notes: 1. Likelihood  $\chi^2$  test or Fisher's exact probability test will be used for group comparison of qualitative measures.
  - 2. Group t-test or Wilcoxon Rank Sum test will be used for group comparison of quantitative measures.
  - 3. For quantitative measures Q1: 25th quantile Q3: 75th quantile.
  - 4. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.
Table 28 (FAS) Analysis results of evaluation immediately after the filling procedure

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Location of tooth to be evaluated | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| UR | XXX (XX.X%) | XXX (XX.X%) | | |
| UL | XXX (XX.X%) | XXX (XX.X%) | | |
| LL | XXX (XX.X%) | XXX (XX.X%) | | |
| LR | XXX (XX.X%) | XXX (XX.X%) | | |
| Location code of UR tooth to be e | valuated | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 11 | XXX (XX.X%) | XXX (XX.X%) | | |
| 12 | XXX (XX.X%) | XXX (XX.X%) | | |
| 13 | XXX (XX.X%) | XXX (XX.X%) | | |
| 14 | XXX (XX.X%) | XXX (XX.X%) | | |
| 15 | XXX (XX.X%) | XXX (XX.X%) | | |
| 16 | XXX (XX.X%) | XXX (XX.X%) | | |
| 17 | XXX (XX.X%) | XXX (XX.X%) | | |
| 18 | XXX (XX.X%) | XXX (XX.X%) | | |
| Location code of UL tooth to be e | valuated | , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 21 | XXX (XX.X%) | XXX (XX.X%) | | |
| 22 | XXX (XX.X%) | XXX (XX.X%) | | |
| 23 | XXX (XX.X%) | XXX (XX.X%) | | |
| 24 | XXX (XX.X%) | XXX (XX.X%) | | |
| 25 | XXX (XX.X%) | XXX (XX.X%) | | |
| 26 | XXX (XX.X%) | XXX (XX.X%) | | |
| 27 | XXX (XX.X%) | XXX (XX.X%) | | |
| 28 | XXX (XX.X%) | XXX (XX.X%) | | |

Notes: 1. Likelihood  $\chi 2$  test or Fisher's exact probability test will be used for group comparison of qualitative measures. 2. Treatment group:  $3M^{TM}$  Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group:  $3M^{TM}$  Filtek<sup>TM</sup> Z350XT.

Table 28 (FAS) Analysis results of evaluation immediately after the filling procedure (cont.)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Location code of LL tooth to | Location code of LL tooth to be evaluated | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 31 | XXX (XX.X%) | XXX (XX.X%) | | |
| 32 | XXX (XX.X%) | XXX (XX.X%) | | |
| 33 | XXX (XX.X%) | XXX (XX.X%) | | |
| 34 | XXX (XX.X%) | XXX (XX.X%) | | |
| 35 | XXX (XX.X%) | XXX (XX.X%) | | |
| 36 | XXX (XX.X%) | XXX (XX.X%) | | |
| 37 | XXX (XX.X%) | XXX (XX.X%) | | |
| 38 | XXX (XX.X%) | XXX (XX.X%) | | |
| Location code of LR tooth to | ` , | , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 41 | XXX (XX.X%) | , , | | |
| 42 | XXX (XX.X%) | , , | | |
| 43 | XXX (XX.X%) | , , | | |
| 44 | XXX (XX.X%) | | | |
| 45 | XXX (XX.X%) | , | | |
| 46 | XXX (XX.X%) | | | |
| 47 | XXX (XX.X%) | , , | | |
| 48 | XXX (XX.X%) | XXX (XX.X%) | | |
| Cavity classification | , | , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Class I cavities | XXX (XX.X%) | , , | | |
| Class II cavities | XXX (XX.X%) | XXX (XX.X%) | | |

Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures. 2. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 29 (FAS) Analysis results of consistency evaluation immediately after the filling procedure

| Measure | es | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|---|
| Retention | n and fractures of the filling | | | | |
| | ses (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| | No marginal fractures of the | , | , | | |
| | filling | XXX (XX.X%) | XXX (XX.X%) | | |
| В. | Minor marginal fractures of the | | | | |
| | filling without exposed dentin, | 7/7/7/ (7/7/ 7/0/) | 3/3/3/ (3/3/ 3/0/) | | |
| C | clinically acceptable; | XXX (XX.X%) | XXX (XX.X%) | | |
| C. | Marginal fractures of the filling with exposed dentin, clinically | | | | |
| | unacceptable | XXX (XX.X%) | XXX (XX.X%) | | |
| NA | | XXX (XX.X%) | XXX (XX.X%) | | |
| | fractures of the filling | 70.01 (70.11770) | 7221 (7212170) | | |
| | ses (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| | No marginal fractures of the | , | , | | |
| | filling | XXX (XX.X%) | XXX (XX.X%) | | |
| B. | Minor marginal fractures of the | | | | |
| | filling without exposed dentin, | | | | |
| _ | clinically acceptable; | XXX (XX.X%) | XXX (XX.X%) | | |
| C. | Marginal fractures of the filling | | | | |
| | with exposed dentin, clinically | VVV (VV V0/) | 3/3/3/ (3/3/ 3/0/) | | |
| NA | unacceptable | XXX (XX.X%) | XXX (XX.X%) | | |
| | and marginal adaptation | XXX (XX.X%) | XXX (XX.X%) | | |
| | ses (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| | Intact contour and continuous | 7011 (7011) | 7221 (7221) | 71.71717171 | 71.71717171 |
| | probing between the filling and | | | | |
| | tooth | XXX (XX.X%) | XXX (XX.X%) | | |
| В. | Pits on the surface of the filling | | | | |
| | and discontinuous probing | | | | |
| | between the filling and tooth | | | | |
| ~ | without exposed dentin; | XXX (XX.X%) | XXX (XX.X%) | | |
| C. | Severe attrition and dents on the | | | | |
| | surface of the filling with exposed dentin, or probes | | | | |
| | hooked at the margins of the | | | | |
| | filling | XXX (XX.X%) | XXX (XX.X%) | | |
| NA | = | XXX (XX.X%) | XXX (XX.X%) | | |
| Proximal | | , , | , , | | |
| | ses (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| | Firm proximal contact | XXX (XX.X%) | XXX (XX.X%) | | |
| В. | Proximal contact is clinically | | | | |
| ~ | acceptable | XXX (XX.X%) | XXX (XX.X%) | | |
| | No proximal contact | XXX (XX.X%) | XXX (XX.X%) | | |
| NA<br>Color ma | | XXX (XX.X%) | XXX (XX.X%) | | |
| | ses (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| | Matching color and transparency | ΛΛΛ (ΛΛΛ) | ΛΛΛ (ΛΛΛ) | Λ.ΛΛΛΛ | Λ.ΛΛΛΛ |
| A. | between the filling and adjacent | | | | |
| | tooth tissues | XXX (XX.X%) | XXX (XX.X%) | | |
| В. | Pits on the surface of the filling | 11111 (11111179) | 11111 (11111179) | | |
| | and discontinuous probing | | | | |
| | between the filling and tooth | | | | |
| | without exposed dentin; | XXX (XX.X%) | XXX (XX.X%) | | |
| C. | Severe attrition and dents on the | | | | |
| | surface of the filling with | | | | |
| | exposed dentin, or probes | | | | |
| | hooked at the margins of the | VVV (VV V0/) | VVV (VV V0/) | | |
| NA | filling | XXX (XX.X%)<br>XXX (XX.X%) | XXX (XX.X%) | | |
| INA | | $\Lambda\Lambda\Lambda$ ( $\Lambda\Lambda.\Lambda$ 70) | XXX (XX.X%) | | |

<sup>2.</sup> Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 29 (FAS) Analysis results of consistency evaluation immediately after the filling procedure (cont.)

| Measure | | Treatment group | | | P value |
|---|---|---|---|---|---|
| Surface re | oughness | | | | |
| | es (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| | After air drying, the surface of | , | , | | |
| | the filling is smooth with luster | | | | |
| | and matching with surrounding | | | | |
| | tooth tissues | XXX (XX.X%) | XXX (XX.X%) | | |
| В. | After air drying, the surface of the | | | | |
| | filling is smooth without luster | XXX (XX.X%) | XXX (XX.X%) | | |
| C. | After air drying, the surface of | | | | |
| | the filling is rough with defects | XXX (XX.X%) | XXX (XX.X%) | | |
| NA<br>C. C | | XXX (XX.X%) | XXX (XX.X%) | | |
| Surface s | | VVV (VVV) | VVV (VVV) | VVVVV | V VVVV |
| | es (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| A. | No staining on the surface of the filling | VVV (VV V0/.) | VVV (VV V%) | | |
| D | Abnormal staining on the surface | XXX (XX.X%) | XXX (XX.X%) | | |
| Б. | of the filling | XXX (XX.X%) | XXX (XX.X%) | | |
| NA | | XXX (XX.X%) | XXX (XX.X%) | | |
| | scoloration and secondary caries | 7221 (721.7170) | 7222 (7212770) | | |
| | es (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| | No discoloration at the interface | () | () | | |
| | between the filling and tooth | XXX (XX.X%) | XXX (XX.X%) | | |
| В. | Partial discoloration at the | , | , | | |
| | interface between the filling and | | | | |
| | tooth, but not extending to pulp | | | | |
| | and removable by polishing; | XXX (XX.X%) | XXX (XX.X%) | | |
| C. | Partial discoloration at the | | | | |
| | interface between the filling and | | | | |
| | tooth extending to pulp and not | | | | |
| | removable by polishing, or | | | | |
| | secondary caries | XXX (XX.X%) | XXX (XX.X%) | | |
| NA | | XXX (XX.X%) | XXX (XX.X%) | | |
| Secondar | | 3/3/3/ (3/3/3/) | 3/3/3/ (3/3/3/) | 37. 37373737 | 37 37373737 |
| | es (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| A. | No discoloration at the interface | VVV (VV V0/) | VVV (VV V0/) | | |
| D | between the filling and tooth Partial discoloration at the | XXX (XX.X%) | XXX (XX.X%) | | |
| Б. | interface between the filling and | | | | |
| | tooth, but not extending to pulp | | | | |
| | and removable by polishing; | XXX (XX.X%) | XXX (XX.X%) | | |
| C | Partial discoloration at the | 7277 (727.7470) | AAA (AA.A70) | | |
| ٠. | interface between the filling and | | | | |
| | tooth extending to pulp and not | | | | |
| | removable by polishing, or | | | | |
| | secondary caries | XXX (XX.X%) | XXX (XX.X%) | | |
| NA | | XXX (XX.X%) | XXX (XX.X%) | | |
| Pulp statu | us | , | , | | |
| Cas | es (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| A. | Normal (temperature test) | XXX (XX.X%) | XXX (XX.X%) | | |
| B. | Temporarily sensitive | | | | |
| | (temperature test) | XXX (XX.X%) | XXX (XX.X%) | | |
| C. | Sensitive and continuous pain, or | | | | |
| | delayed pain (temperature test) | XXX (XX.X%) | XXX (XX.X%) | | |
| D. | No response (electric pulp testing) | | XXX (XX.X%) | | |
| NA | | XXX (XX.X%) | XXX (XX.X%) | | |

Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures. 2. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 30 (FAS) The analysis results of primary efficacy measure - clinical acceptance rate of the filling at the 1 year follow-up visit after the filling procedure

| Measures | Treatment group | Control grou | p Statistics | P value |
|---|---|---|---|---|
| Clinical acceptance rate of | the filling at the 1 year follow-up | visit after the | filling procedure | <b>,</b> #1 |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Acceptable | XXX (XX.X%) | XXX (XX.Xº | %) | |
| Not acceptable | XXX (XX.X%) | XXX (XX.Xº | %) | |
| Clinical acceptance rate of | the filling at the 1 year follow-up | visit after the | filling procedure | #2 |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | | |
| Acceptable | XXX (XX.X%) | XXX (XX.Xº | %) | |
| Not acceptable | XXX (XX.X%) | XXX (XX.Xº | %) | |
| | Difference in acceptance | rate XX.X | % [XX.X%; X | X.X%] |
| | (treatment - control) and 95% | | _ | - |
| | p value of non-inferiority | test X.XX | XX | |
| Clinical acceptance rate of | the filling at the 1 year follow-up | visit after the | filling procedure | #3 |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | | |
| Acceptable | XXX (XX.X%) | XXX (XX.Xº | %) | |
| Not acceptable | XXX (XX.X%) | XXX (XX.Xº | %) | |
| | Difference in acceptance | rate XX.X | % [XX.X%; X | X.X%] |
| | (treatment - control) and 95% | | . , | , |
| | p value of non-inferiority | test X.XX | XX | |

- Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures.
  - 2. #2: Analyze with CMH Chi square test adjusted for center effect;
  - 3. #1: Primary efficacy measures of subjects who are lost to follow-up will not be processed;
    - #2: Primary efficacy measures of subjects who are lost to follow-up will not be acceptable for carry forward;
    - #3: Primary efficacy measures of subjects who are lost to follow-up will be carried forward by last follow-up
  - 4. The definition of clinically acceptable filling at the 1 year follow-up visit is: grade A for retention and fracture of the filling 1 year after the filling procedure; grade A or B for marginal fracture, contour and marginal adaptation of the filling.
  - 5. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.
  - 6. Borderline value of noninferiority is set to 7%.

Table 31 (FAS) The analysis results of primary efficacy measure - clinical acceptance rate of the filling at the 1 year follow-up visit after the filling procedure (Tipping Point analysis results)

| Suppleme | nt of subjects | who are lost to | follow-up | | Clinical acce | eptance rate | | 7.00 |
|---|---|---|---|---|---|---|---|---|
| Treatment group | | Contro | ol group | Treatment group | | Control group | | Difference in acceptance rate # (treatment - control) and |
| Acceptable | Not acceptable | Acceptable | Not acceptable | Acceptable | Not acceptable | Acceptable | Not acceptable | 95% CI |
| XXX | XXX | XXX | XXX | XX.X (XX.X%) | XX.X (XX.X%) | XX.X (XX.X%) | XX.X (XX.X%) | XX.X% [XX.X%; XX.X%] |
| | | | | | •••• | | | ••••• |

- 2. #: Analyze with CMH Chi square test adjusted for center effect;
- 3. The definition of clinically acceptable filling at the 1 year follow-up visit is: grade A for retention and fracture of the filling 1 year after the filling procedure; grade A or B for marginal fracture, contour and marginal adaptation of the filling.

  4. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.
- 5. Borderline value of noninferiority is set to 7%.

Table 32 (FAS) The analysis results of primary efficacy measure - clinical acceptance rate of the filling at the 1 year follow-up visit after the filling procedure (subgroup analysis of each center)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Clinical acceptance rate of the filling at the 1 year follow-up visit after the filling procedure at Peking | | | | |
| University Hospital of Stomatology | | | | |
| Cases (Nmiss) | XXX(XXX) | XXX(XXX) | X.XXXX | X.XXXX |
| Acceptable | XXX (XX.X%) | XXX (XX.X%) | | |
| Not acceptable | XXX (XX.X%) | XXX (XX.X%) | | |
| Clinical acceptance rate of the filling at the 1 year follow-up visit after the filling procedure at Hospital | | | | |
| of Stomatology Wuhan University | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Acceptable | XXX (XX.X%) | XXX (XX.X%) | | |
| Not acceptable | XXX (XX.X%) | XXX (XX.X%) | | |
| Clinical acceptance rate of the filling at th | e 1 year follow-up | visit after the filling | ng procedure | at Beijing |
| Stomatological Hospital Capital Medical Un | iversity | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Acceptable | XXX (XX.X%) | XXX (XX.X%) | | |
| Not acceptable | XXX (XX.X%) | XXX (XX.X%) | | |

- 2. The definition of clinically acceptable filling at the 1 year follow-up visit is: grade A for retention and fracture of the filling 1 year after the filling procedure; grade A or B for marginal fracture, contour and marginal adaptation of the filling.
- 3. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.
- 4. Borderline value of noninferiority is set to 7%.

Table 33 (PPS) The analysis results of primary efficacy measure - clinical acceptance rate of the filling at the 1 year follow-up visit after the filling procedure

| Measures | Treatment group Control group |
|---|---|
| | filling at the 1 year follow-up visit after the filling procedure# |
| Cases (Nmiss) | XXX(XXX) $XXX(XXX)$ |
| Acceptable | XXX (XX.X%) XXX (XX.X%) |
| Not acceptable | XXX (XX.X%) XXX (XX.X%) |
| <del></del> | Difference in acceptance rate XX.X% [XX.X%; XX.X%] |
| | (treatment - control) and 95% CI |
| | p value of non-inferiority test X.XXXX |

- 2. #: Analyze with CMH Chi square test adjusted for center effect;
- 3. The definition of clinically acceptable filling at the 1 year follow-up visit is: grade A for retention and fracture of the filling 1 year after the filling procedure; grade A or B for marginal fracture, contour and marginal adaptation of the filling.
- Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.
- 5. Borderline value of noninferiority is set to 7%.

Table 34 (PPS) The analysis results of primary efficacy measure - clinical acceptance rate of the filling at the 1 year follow-up visit after the filling procedure (subgroup analysis of each center)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Clinical acceptance rate of the filling at the 1 year follow-up visit after the filling procedure at Peking | | | | |
| University Hospital of Stomatology | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Acceptable | XXX (XX.X%) | XXX (XX.X%) | | |
| Not acceptable | XXX (XX.X%) | XXX (XX.X%) | | |
| Clinical acceptance rate of the filling at the 1 | Clinical acceptance rate of the filling at the 1 year follow-up visit after the filling procedure at Hospital of | | | |
| Stomatology Wuhan University | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Acceptable | XXX (XX.X%) | XXX (XX.X%) | | |
| Not acceptable | XXX (XX.X%) | XXX (XX.X%) | | |
| Clinical acceptance rate of the filling at the 1 | year follow-up vi | sit after the filling | procedure at | Beijing |
| Stomatological Hospital Capital Medical Un | iversity | | - | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Acceptable | XXX (XX.X%) | XXX (XX.X%) | | |
| Not acceptable | XXX (XX.X%) | XXX (XX.X%) | | |

- 2. The definition of clinically acceptable filling at the 1 year follow-up visit is: grade A for retention and fracture of the filling 1 year after the filling procedure; grade A or B for marginal fracture, contour and marginal adaptation of the filling.
- 3. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.
- 4. Borderline value of noninferiority is set to 7%.

Table 35 (FAS) The analysis results of secondary efficacy measure - clinical acceptance rate of the filling at the 1 week follow-up visit after the filling procedure

| at the 1 week lone, up visit after the many procedure | | | |
|---|---|---|---|
| Treatment group | Control group | Statistics | P value |
| XXX (XXX)<br>XXX (XX.X%) | XXX (XXX)<br>XXX (XX.X%) | procedure | |
| XXX (XX.X%) | XXX(XX.X%) | | |
| | Treatment group week follow-up vi XXX (XXX) XXX (XX.X%) | Treatment group Control group | Treatment group Control group Statistics week follow-up visit after the filling procedure XXX (XXX) XXX (XXX) XXX (XXXX) XXX (XXXX) |

- Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures.
  - 2. #: Analyze with CMH Chi square test adjusted for center effect;
  - 3. The definition of clinically acceptable filling at the 1 week follow-up is: grade A or B 1 week after the filling procedure for all the measures, including retention and fracture of the filling, marginal fracture, contour and marginal adaptation, proximal contact, color match, surface roughness, surface staining, marginal discoloration, secondary caries and pulp status;
  - 4. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 36 (FAS) The analysis results of secondary efficacy measures for evaluation - proximal contact, color match, surface roughness, surface staining, marginal discoloration, secondary caries

| and pulp status | vear after the f | illing procedure |
|-----------------|------------------|------------------|
|-----------------|------------------|------------------|

| | X | | | |
|---|---|---|---|---|
| Measures | Treatment group | Control group | Statistics | P value |
| Proximal contact | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| <ul> <li>A. Firm proximal contact</li> </ul> | XXX (XX.X%) | XXX (XX.X%) | | |
| B. Proximal contact is clinically | | | | |
| acceptable | XXX (XX.X%) | XXX (XX.X%) | | |
| <ul><li>C. No proximal contact</li></ul> | XXX (XX.X%) | XXX (XX.X%) | | |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |
| Color match | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| A. Matching color and transparency between the filling and adjacent | | | | |
| tooth tissues | XXX (XX.X%) | XXX (XX.X%) | | |
| B. Pits on the surface of the filling and discontinuous probing | | | | |
| between the filling and tooth | VVV (VV V0/) | VVV (VV V0/) | | |
| without exposed dentin C. Severe attrition and dents on the | XXX (XX.X%) | XXX (XX.X%) | | |
| surface of the filling with | | | | |
| exposed dentin, or probes | | | | |
| hooked at the margins of the | VVV (VV V0/) | VVV (VV V0/) | | |
| filling | XXX (XX.X%) | XXX (XX.X%) | | |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |
| Surface roughness<br>Cases (Nmiss) | VVV (VVV) | VVV (VVV) | vvvvv | v vvvv |
| , | XXX (XXX) | XXX (XXX) | Λ.ΛΛΛΛ | X.XXXX |
| A. After air drying, the surface of the filling is smooth with luster | | | | |
| and matching with surrounding | VVV (VV V0/) | VVV (VV V0/) | | |
| tooth tissues | XXX (XX.X%) | XXX (XX.X%) | | |
| B. After air drying, the surface of | | | | |
| the filling is smooth without | 3/3/3/ (3/3/ 3/0/) | 3/3/3/ (3/3/ 3/0/) | | |
| luster | XXX (XX.X%) | XXX (XX.X%) | | |
| C. After air drying, the surface of | | | | |
| the filling is rough with defects | XXX (XX.X%) | XXX (XX.X%) | | |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |
| Surface staining | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| A. No staining on the surface of the | | | | |
| filling | XXX (XX.X%) | XXX (XX.X%) | | |
| B. Abnormal staining on the surface | | | | |
| of the filling | XXX (XX.X%) | XXX (XX.X%) | | |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |
| Marginal discoloration and secondary caries | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| A. No discoloration at the interface | | | | |
| between the filling and tooth | XXX (XX.X%) | XXX (XX.X%) | | |
| B. Partial discoloration at the | | | | |
| interface between the filling and | | | | |
| tooth, but not extending to pulp | | | | |
| and removable by polishing | XXX (XX.X%) | XXX (XX.X%) | | |
| C. Partial discoloration at the | , , | , | | |
| interface between the filling and | | | | |
| tooth extending to pulp and not | | | | |
| removable by polishing, or | | | | |
| secondary caries | XXX (XX.X%) | XXX (XX.X%) | | |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |
| 1117 | 11111 (1111.7170) | 212121 (2121.21/0) | | |

| Seconda | ry caries | | | | |
|---|---|---|---|---|---|
| Cas | ses (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| A. | No discoloration at the interface | | | | |
| | between the filling and tooth | XXX (XX.X%) | XXX (XX.X%) | | |
| B. | Partial discoloration at the | | | | |
| | interface between the filling and | | | | |
| | tooth, but not extending to pulp | | | | |
| | and removable by polishing | XXX (XX.X%) | XXX (XX.X%) | | |
| C. | Partial discoloration at the | | | | |
| | interface between the filling and | | | | |
| | tooth extending to pulp and not | | | | |
| | removable by polishing, or | | | | |
| | secondary caries | XXX (XX.X%) | XXX (XX.X%) | | |
| NA | <u>.</u> | XXX (XX.X%) | XXX (XX.X%) | | |

Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures.

2. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 36 (FAS) The analysis results of secondary efficacy measures - proximal contact, color match, surface roughness, surface staining, marginal discoloration, secondary caries and pulp status 1 year after the filling procedure (cont.)

| Measur | es | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|---|
| Pulp sta | itus | | | | |
| Cas | ses (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| A. | Normal (temperature test) | XXX (XX.X%) | XXX (XX.X%) | | |
| B. | Temporarily sensitive | , | ` , | | |
| | (temperature test) | XXX (XX.X%) | XXX (XX.X%) | | |
| C. | Sensitive and continuous | , | , | | |
| | pain, or delayed pain | | | | |
| | (temperature test) | XXX (XX.X%) | XXX (XX.X%) | | |
| D. | No response (electric pulp | | | | |
| | testing) | XXX (XX.X%) | XXX (XX.X%) | | |
| NA | | XXX (XX.X%) | XXX (XX.X%) | | |

Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative measures.

2. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 37 (FAS) Analysis results of oral soft tissue examination at the 1 week (± 3 days) follow-up visit after the filling procedure

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Conduct oral soft tissue examina | ation | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Normality of oral soft tissue | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Oral soft tissue area | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 1 | XXX (XX.X%) | XXX (XX.X%) | | |
| 2 | XXX (XX.X%) | XXX (XX.X%) | | |
| | XXX (XX.X%) | XXX (XX.X%) | | |
| Size a (mm) of oral examination | result (area level) | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| $Mean \pm SD$ | $XX.XX\pm XX.XX$ | $XX.XX\pm XX.XX$ | | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Size b (mm) of oral examination | , | , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Mean $\pm$ SD | XX.XX±XX.XX | XX.XX±XX.XX | 11111111111 | |
| Median | XX.XX | XX.XX | | |
| Q1; Q3 | XX.XX; XX.XX | | | |
| Minimum; Maximum | XX.XX; XX.XX | XX.XX; XX.XX | | |
| Size a*b (mm) of oral examination | , | | | |
| XX*XX | XXX (XX.X%) | XXX (XX.X%) | | |
| ΑΛ ΑΛ | XXX (XX.X%) $XXX (XX.X%)$ | XXX (XX.X%) $XXX (XX.X%)$ | | |
| <br>Clinical significance of oral exa | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | | <i>A.A.</i> | / <b>1./1/1/1</b> / |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |

<sup>2.</sup> Group t-test or Wilcoxon Rank Sum test will be used for group comparison of quantitative measures.

<sup>3.</sup> For quantitative measures, Q1: 25th quantile; Q3: 75th quantile

<sup>4.</sup> Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 37 (FAS) Analysis results of oral soft tissue examination at the 1 week (± 3 days) follow-up visit after the filling procedure (cont.)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Examination results area (area level) | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| None | XXX (XX.X%) | XXX (XX.X%) | | |
| 1 | XXX (XX.X%) | XXX (XX.X%) | | |
| 2 | XXX (XX.X%) | XXX (XX.X%) | | |
| 3 | XXX (XX.X%) | XXX (XX.X%) | | |
| 4 | XXX (XX.X%) | XXX (XX.X%) | | |
| 5 | XXX (XX.X%) | XXX (XX.X%) | | |
| 6 | XXX (XX.X%) | XXX (XX.X%) | | |
| 7 | XXX (XX.X%) | XXX (XX.X%) | | |
| 8 | XXX (XX.X%) | XXX (XX.X%) | | |
| 9 | XXX (XX.X%) | XXX (XX.X%) | | |
| 10 | XXX (XX.X%) | XXX (XX.X%) | | |
| 11 | XXX (XX.X%) | XXX (XX.X%) | | |
| 12 | XXX (XX.X%) | XXX (XX.X%) | | |
| 13 | XXX (XX.X%) | XXX (XX.X%) | | |
| 14 | XXX (XX.X%) | XXX (XX.X%) | | |
| 15 | XXX (XX.X%) | XXX (XX.X%) | | |
| 16 | XXX (XX.X%) | XXX (XX.X%) | | |
| 17 | XXX (XX.X%) | XXX (XX.X%) | | |
| 18 | XXX (XX.X%) | XXX (XX.X%) | | |
| 19 | XXX (XX.X%) | XXX (XX.X%) | | |
| 20 | XXX (XX.X%) | XXX (XX.X%) | | |
| 21 | XXX (XX.X%) | XXX (XX.X%) | | |
| 22 | XXX (XX.X%) | XXX (XX.X%) | | |
| 23 Dorsum linguae | XXX (XX.X%) | XXX (XX.X%) | | |
| 24 Ventral linguae | XXX (XX.X%) | XXX (XX.X%) | | |
| 25 Apex linguae | XXX (XX.X%) | XXX (XX.X%) | | |
| 26 Lingual margin | XXX (XX.X%) | XXX (XX.X%) | | |
| 27 Tongue base | XXX (XX.X%) | XXX (XX.X%) | | |
| 28 Epiglottis | XXX (XX.X%) | XXX (XX.X%) | | |

- 2. Group t-test or Wilcoxon Rank Sum test will be used for group comparison of quantitative measures.
- 3. For quantitative measures, Q1: 25th quantile; Q3: 75th quantile
   4. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 38 (FAS) Analysis results of filling treatment and digital photos at the 1 week (± 3 days) follow-up visit after the filling procedure

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Filling needs treatment | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Take digital photos | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos | | | | |
| Photos of occlusal surface | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos | , | , | | |
| Photos of occlusal surface (with occlusa | al contacts marked) | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos | , | , | | |
| Photos of median occlusion | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos | , | , | | |
| Photos of antagonist tooth | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos | , | , | | |
| Photos of buccal surface | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos | , | , | | |
| Photos of lingual surface | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | · <b>-</b> | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos | (1212117) | (-222273) | | |
| Other | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |

Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative

<sup>2.</sup> Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 39 (FAS) Analysis results of evaluation results at the 1 week (± 3 days) follow-up visit after the filling procedure

| | arter the iming p | | | |
|---|---|---|---|---|
| Measures | Treatment group | Control group | Statistics | P value |
| Location of tooth to be evaluated | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| UR | XXX (XX.X%) | XXX (XX.X%) | | |
| UL | XXX (XX.X%) | XXX (XX.X%) | | |
| LL | XXX (XX.X%) | XXX (XX.X%) | | |
| LR | XXX (XX.X%) | XXX (XX.X%) | | |
| Location code of UR tooth to be | evaluated | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 11 | XXX (XX.X%) | XXX (XX.X%) | | |
| 12 | XXX (XX.X%) | XXX (XX.X%) | | |
| 13 | XXX (XX.X%) | XXX (XX.X%) | | |
| 14 | XXX (XX.X%) | XXX (XX.X%) | | |
| 15 | XXX (XX.X%) | XXX (XX.X%) | | |
| 16 | XXX (XX.X%) | XXX (XX.X%) | | |
| 17 | XXX (XX.X%) | | | |
| 18 | XXX (XX.X%) | | | |
| Location code of UL tooth to be e | valuated | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 21 | XXX (XX.X%) | XXX (XX.X%) | | |
| 22 | XXX (XX.X%) | XXX (XX.X%) | | |
| 23 | XXX (XX.X%) | | | |
| 24 | XXX (XX.X%) | XXX (XX.X%) | | |
| 25 | XXX (XX.X%) | XXX (XX.X%) | | |
| 26 | XXX (XX.X%) | XXX (XX.X%) | | |
| 27 | XXX (XX.X%) | , , | | |
| 28 | XXX (XX.X%) | XXX (XX.X%) | | |

- Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative
  - 2. Treatment group:  $3M^{TM}$  Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group:  $3M^{TM}$  Filtek<sup>TM</sup> Z350XT.

Table 39 (FAS) Analysis results of evaluation results at the 1 week ( $\pm$  3 days) follow-up visit after the filling procedure (cont.)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Location code of LL tooth to be | e evaluated | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 31 | XXX (XX.X%) | XXX (XX.X%) | | |
| 32 | XXX (XX.X%) | XXX (XX.X%) | | |
| 33 | XXX (XX.X%) | XXX (XX.X%) | | |
| 34 | XXX (XX.X%) | XXX (XX.X%) | | |
| 35 | XXX (XX.X%) | | | |
| 36 | XXX (XX.X%) | XXX (XX.X%) | | |
| 37 | XXX (XX.X%) | XXX (XX.X%) | | |
| 38 | XXX (XX.X%) | | | |
| Location code of LR tooth to be | * | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 41 | XXX (XX.X%) | XXX (XX.X%) | | |
| 42 | XXX (XX.X%) | XXX (XX.X%) | | |
| 43 | XXX (XX.X%) | XXX (XX.X%) | | |
| 44 | XXX (XX.X%) | XXX (XX.X%) | | |
| 45 | XXX (XX.X%) | XXX (XX.X%) | | |
| 46 | XXX (XX.X%) | XXX (XX.X%) | | |
| 47 | XXX (XX.X%) | XXX (XX.X%) | | |
| 48 | XXX (XX.X%) | XXX (XX.X%) | | |
| Cavity classification | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Class I cavities | XXX (XX.X%) | | | |
| Class II cavities | XXX (XX.X%) | XXX (XX.X%) | | |

<sup>2.</sup> Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 40 (FAS) Analysis results of consistency evaluation results at the 1 week ( $\pm$  3 days) follow-up visit after the filling procedure

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Retention and fractures of the filling | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| A. No marginal fractures of the | | | | |
| filling | XXX (XX.X%) | XXX (XX.X%) | | |
| B. Minor marginal fractures of | | | | |
| the filling without exposed | 3/3/3/ (3/3/ 3/0/) | 373737 (3737 370/) | | |
| dentin, clinically acceptable; | XXX (XX.X%) | XXX (XX.X%) | | |
| C. Marginal fractures of the filling with exposed dentin, | | | | |
| clinically unacceptable | XXX (XX.X%) | XXX (XX.X%) | | |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |
| Marginal fractures of the filling | 11111 (11111170) | 11111 (11111170) | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| A. No marginal fractures of the | , , | | | |
| filling | XXX (XX.X%) | XXX (XX.X%) | | |
| B. Minor marginal fractures of | | | | |
| the filling without exposed | 77777 (7777 770 () | ****** (**** **** (*) | | |
| dentin, clinically acceptable; | XXX (XX.X%) | XXX (XX.X%) | | |
| C. Marginal fractures of the filling with exposed dentin, | | | | |
| clinically unacceptable | XXX (XX.X%) | XXX (XX.X%) | | |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |
| Contour and marginal adaptation | 1221 (1221173) | 11111 (11111173) | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| A. Intact contour and continuous | | | | |
| probing between the filling | | | | |
| and tooth | XXX (XX.X%) | XXX (XX.X%) | | |
| B. Pits on the surface of the | | | | |
| filling and discontinuous probing between the filling | | | | |
| and tooth without exposed | | | | |
| dentin; | XXX (XX.X%) | XXX (XX.X%) | | |
| C. Severe attrition and dents on | 1222 (122270) | 11111 (11111170) | | |
| the surface of the filling with | | | | |
| exposed dentin, or probes | | | | |
| hooked at the margins of the | | | | |
| filling | XXX (XX.X%) | XXX (XX.X%) | | |
| NA<br>D | XXX (XX.X%) | XXX (XX.X%) | | |
| Proximal contact | VVV (VVV) | VVV (VVV) | vvvvv | vvvvv |
| Cases (Nmiss) A. Firm proximal contact | XXX (XXX)<br>XXX (XX.X%) | XXX (XXX)<br>XXX (XX.X%) | X.XXXX | X.XXXX |
| B. Proximal contact is clinically | $\Lambda\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda/0)$ | $\Lambda\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda/0)$ | | |
| acceptable | XXX (XX.X%) | XXX (XX.X%) | | |
| r | | , , | | |
| <ul><li>C. No proximal contact</li></ul> | XXX (XX.X%) | XXX (XX.X%) | | |

| Color match | | | | |
|---|---|---|---|---|
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| A. Matching color and transparency between the filling and adjacent tooth | | | | |
| tissues | XXX (XX.X%) | XXX (XX.X%) | | |
| B. Pits on the surface of the filling and discontinuous probing between the filling and tooth without exposed | | | | |
| dentin; | XXX (XX.X%) | XXX (XX.X%) | | |
| C. Severe attrition and dents on<br>the surface of the filling with<br>exposed dentin, or probes<br>hooked at the margins of the | | | | |
| filling | XXX (XX.X%) | XXX (XX.X%) | | |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |

- Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative
  - 2. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 41 (FAS) Analysis results of consistency evaluation results at the 1 week (± 3 days) follow-up visit after the filling procedure (cont.)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Surface roughness | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| A. After air drying, the surface of | | | | |
| the filling is smooth with | | | | |
| luster and matching with surrounding tooth tissues | XXX (XX.X%) | XXX (XX.X%) | | |
| B. After air drying, the surface of | $\Lambda\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda/0)$ | AAA(AA.A/0) | | |
| the filling is smooth without | | | | |
| luster | XXX (XX.X%) | XXX (XX.X%) | | |
| C. After air drying, the surface of | | | | |
| the filling is rough with | ************************************** | <b>373737</b> (3737 370 () | | |
| defects | XXX (XX.X%) | XXX (XX.X%) | | |
| NA<br>Surface staining | XXX (XX.X%) | XXX (XX.X%) | | |
| Surface staining Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| A. No staining on the surface of | $\Lambda\Lambda\Lambda$ $(\Lambda\Lambda\Lambda)$ | ΑΛΛ (ΛΛΛ) | Α.ΑΑΑΑ | Λ.ΛΛΛΛ |
| the filling | XXX (XX.X%) | XXX (XX.X%) | | |
| B. Abnormal staining on the | , | , | | |
| surface of the filling | XXX (XX.X%) | XXX (XX.X%) | | |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |
| Marginal discoloration and secondary cari | | 3/3/3/ (3/3/3/) | 37 37373737 | 37. 37373737 |
| Cases (Nmiss) A. No discoloration at the | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| interface between the filling | | | | |
| and tooth | XXX (XX.X%) | XXX (XX.X%) | | |
| B. Partial discoloration at the | , | , | | |
| interface between the filling | | | | |
| and tooth, but not extending | | | | |
| to pulp and removable by polishing; | XXX (XX.X%) | XXX (XX.X%) | | |
| C. Partial discoloration at the | $\Lambda\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda/0)$ | $\Lambda\Lambda\Lambda$ $(\Lambda\Lambda.\Lambda/0)$ | | |
| interface between the filling | | | | |
| and tooth extending to pulp | | | | |
| and not removable by | | | | |
| polishing, or secondary caries | | XXX (XX.X%) | | |
| NA<br>C | XXX (XX.X%) | XXX (XX.X%) | | |
| Secondary caries | VVV (VVV) | VVV (VVV) | X.XXXX | X.XXXX |
| Cases (Nmiss) A. No discoloration at the | XXX (XXX) | XXX (XXX) | Λ.ΛΛΛΛ | Λ.ΛΛΛΛ |
| interface between the filling | | | | |
| and tooth | XXX (XX.X%) | XXX (XX.X%) | | |
| B. Partial discoloration at the | | | | |
| interface between the filling | | | | |
| and tooth, but not extending | | | | |
| to pulp and removable by polishing; | XXX (XX.X%) | XXX (XX.X%) | | |
| C. Partial discoloration at the | 71.71 (71.71.71) | 7474 (7474.7470) | | |
| interface between the filling | | | | |
| and tooth extending to pulp | | | | |
| and not removable by | | | | |
| polishing, or secondary caries | XXX (XX.X%) | XXX (XX.X%) | | |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |

| Pulp status | | | | |
|---|---|---|---|---|
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| A. Normal (temperature test) | XXX (XX.X%) | XXX (XX.X%) | | |
| B. Temporarily sensitive | | | | |
| (temperature test) | XXX (XX.X%) | XXX (XX.X%) | | |
| C. Sensitive and continuous pain, or delayed pain | | | | |
| (temperature test) | XXX (XX.X%) | XXX (XX.X%) | | |
| D. No response (electric pulp | | | | |
| testing) | XXX (XX.X%) | XXX (XX.X%) | | |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |

<sup>2.</sup> Treatment group:  $3M^{TM}$  Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group:  $3M^{TM}$  Filtek<sup>TM</sup> Z350XT.

Table 42 (FAS) Analysis results of oral soft tissue examination at the 12 months (± 1 month) follow-up visit after the filling procedure

| XX (XX.X%)<br>XX (XX.X%)<br>XX (XXX)<br>XX (XX.X%)<br>XX (XX.X%) | | X.XXXX<br>X.XXXX |
|---|---|---|
| XX (XX.X%)<br>XX (XX.X%)<br>XX (XXX)<br>XX (XX.X%)<br>XX (XX.X%) | | |
| XX (XX.X%)<br>XX (XX.X%)<br>XX (XXX)<br>XX (XX.X%)<br>XX (XX.X%) | | |
| XX (XX.X%) XX (XXX) XX (XX.X%) XX (XX.X%) | X.XXXX | X.XXXX |
| XX (XXX)<br>XX (XX.X%)<br>XX (XX.X%) | X.XXXX | X.XXXX |
| XX (XX.X%)<br>XX (XX.X%) | X.XXXX | X.XXXX |
| XX (XX.X%)<br>XX (XX.X%) | X.XXXX | X.XXXX |
| XX (XX.X%) | | |
| , | | |
| XX (XXX) | | |
| XX(XXX) | | |
| | X.XXXX | X.XXXX |
| XX (XX.X%) | | |
| XX (XX.X%) | | |
| XX (XX.X%) | | |
| , | X.XXXX | X.XXXX |
| $X.XX\pm XX.XX$ | | |
| X.XX | | |
| X.XX; XX.XX | | |
| X.XX; XX.XX | | |
| XX (XXX) | X.XXXX | X.XXXX |
| X.XX±XX.XX | | |
| X.XX | | |
| X.XX; XX.XX | | |
| X.XX; XX.XX | | |
| (X (XX.X%) | | |
| , | | |
| ( | | |
| XX (XXX) | X.XXXX | X.XXXX |
| XX (XX.X%) | | <del>-</del> |
| XX (XX.X%) | | |
| | X (XX.X%) X (XX.X%) X (XXX.X%) X (XXX.XX) .XX±XX.XX .XX; XX.XX | X (XX.X%) X (XX.X%) X (XXXX) X (XXXX) X (XXXX) X (XXXX XX; XX.XX |

- 2. Group t-test or Wilcoxon Rank Sum test will be used for group comparison of quantitative measures.
- 3. For quantitative measures, Q1: 25th quantile; Q3: 75th quantile
- 4. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 42 (FAS) Analysis results of oral soft tissue examination at the 12 months (± 1 month) follow-up visit after the filling procedure (cont.)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Examination results area (area level) | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| None | XXX (XX.X%) | XXX (XX.X%) | | |
| 1 | XXX (XX.X%) | XXX (XX.X%) | | |
| 2 | XXX (XX.X%) | XXX (XX.X%) | | |
| 3 | XXX (XX.X%) | XXX (XX.X%) | | |
| 4 | XXX (XX.X%) | XXX (XX.X%) | | |
| 5 | XXX (XX.X%) | XXX (XX.X%) | | |
| 6 | XXX (XX.X%) | XXX (XX.X%) | | |
| 7 | XXX (XX.X%) | XXX (XX.X%) | | |
| 8 | XXX (XX.X%) | XXX (XX.X%) | | |
| 9 | XXX (XX.X%) | XXX (XX.X%) | | |
| 10 | XXX (XX.X%) | XXX (XX.X%) | | |
| 11 | XXX (XX.X%) | XXX (XX.X%) | | |
| 12 | XXX (XX.X%) | XXX (XX.X%) | | |
| 13 | XXX (XX.X%) | XXX (XX.X%) | | |
| 14 | XXX (XX.X%) | XXX (XX.X%) | | |
| 15 | XXX (XX.X%) | XXX (XX.X%) | | |
| 16 | XXX (XX.X%) | XXX (XX.X%) | | |
| 17 | XXX (XX.X%) | XXX (XX.X%) | | |
| 18 | XXX (XX.X%) | XXX (XX.X%) | | |
| 19 | XXX (XX.X%) | XXX (XX.X%) | | |
| 20 | XXX (XX.X%) | XXX (XX.X%) | | |
| 21 | XXX (XX.X%) | XXX (XX.X%) | | |
| 22 | XXX (XX.X%) | XXX (XX.X%) | | |
| 23 Dorsum linguae | XXX (XX.X%) | XXX (XX.X%) | | |
| 24 Ventral linguae | XXX (XX.X%) | XXX (XX.X%) | | |
| 25 Apex linguae | XXX (XX.X%) | XXX (XX.X%) | | |
| 26 Lingual margin | XXX (XX.X%) | XXX (XX.X%) | | |
| 27 Tongue base | XXX (XX.X%) | XXX (XX.X%) | | |
| 28 Epiglottis | XXX (XX.X%) | XXX (XX.X%) | | |

- 2. Group t-test or Wilcoxon Rank Sum test will be used for group comparison of quantitative measures.
- 3. For quantitative measures, Q1: 25th quantile; Q3: 75th quantile
- 4. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 43 (FAS) Analysis results of filling treatment and digital photos at the 12 months (± 1 month) follow-up

visit after the filling procedure

| Measures | 0 1 | Control group | Statistics | P value |
|---|---|---|---|---|
| Filling needs treatment | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Take digital photos | , | ` , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos | | | | |
| Photos of occlusal surface | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos | | | | |
| Photos of occlusal surface (with occl | usal contacts marked) | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos | , | , | | |
| Photos of median occlusion | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos | , | , | | |
| Photos of antagonist tooth | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | , , | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos | , | , | | |
| Photos of buccal surface | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos | ( ) | , | | |
| Photos of lingual surface | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Type of photos | 1111 (111117) | 11111 (11111170) | | |
| Other | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | 1 2.12 22 22 22 2 | 1 2.1. 2.2 2.2 2.2 |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |

<sup>2.</sup> Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 44 (FAS) Analysis results of evaluation results at the 12 months (± 1 month) follow-up visit after the filling procedure

| | ming proced | uuic | | |
|---|---|---|---|---|
| Measures | Treatment group | Control group | Statistics | P value |
| Location of tooth to be evaluated | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| UR | XXX (XX.X%) | XXX (XX.X%) | | |
| UL | XXX (XX.X%) | | | |
| LL | XXX (XX.X%) | XXX (XX.X%) | | |
| LR | XXX (XX.X%) | XXX (XX.X%) | | |
| Location code of UR tooth to be e | valuated | • | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 11 | XXX (XX.X%) | XXX (XX.X%) | | |
| 12 | XXX (XX.X%) | XXX (XX.X%) | | |
| 13 | XXX (XX.X%) | XXX (XX.X%) | | |
| 14 | XXX (XX.X%) | XXX (XX.X%) | | |
| 15 | XXX (XX.X%) | XXX (XX.X%) | | |
| 16 | XXX (XX.X%) | | | |
| 17 | XXX (XX.X%) | XXX (XX.X%) | | |
| 18 | XXX (XX.X%) | XXX (XX.X%) | | |
| Location code of UL tooth to be e | valuated | • | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 21 | XXX (XX.X%) | XXX (XX.X%) | | |
| 22 | XXX (XX.X%) | XXX (XX.X%) | | |
| 23 | XXX (XX.X%) | | | |
| 24 | XXX (XX.X%) | XXX (XX.X%) | | |
| 25 | XXX (XX.X%) | | | |
| 26 | XXX (XX.X%) | | | |
| 27 | XXX (XX.X%) | , | | |
| 28 | XXX (XX.X%) | XXX (XX.X%) | | |

- Notes: 1. Likelihood χ2 test or Fisher's exact probability test will be used for group comparison of qualitative
  - 2. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 44 (FAS) Analysis results of evaluation results at the 12 months (± 1 month) follow-up visit after the filling procedure (cont.)

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| | | e entre i gre up | | |
| Location code of LL tooth to b | e evaluated | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 31 | XXX (XX.X%) | XXX (XX.X%) | | |
| 32 | XXX (XX.X%) | XXX (XX.X%) | | |
| 33 | XXX (XX.X%) | XXX (XX.X%) | | |
| 34 | XXX (XX.X%) | XXX (XX.X%) | | |
| 35 | XXX (XX.X%) | XXX (XX.X%) | | |
| 36 | XXX (XX.X%) | XXX (XX.X%) | | |
| 37 | XXX (XX.X%) | XXX (XX.X%) | | |
| 38 | XXX (XX.X%) | XXX (XX.X%) | | |
| Location code of LR tooth to b | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| 41 | XXX (XX.X%) | XXX (XX.X%) | | |
| 42 | XXX (XX.X%) | XXX (XX.X%) | | |
| 43 | XXX (XX.X%) | XXX (XX.X%) | | |
| 44 | XXX (XX.X%) | XXX (XX.X%) | | |
| 45 | XXX (XX.X%) | XXX (XX.X%) | | |
| 46 | XXX (XX.X%) | XXX (XX.X%) | | |
| 47 | XXX (XX.X%) | XXX (XX.X%) | | |
| 48 | XXX (XX.X%) | XXX (XX.X%) | | |
| Cavity classification | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Class I cavities | XXX (XX.X%) | • • • | | |
| Class II cavities | XXX (XX.X%) | | | |

<sup>2.</sup> Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 45 (FAS) Analysis results of consistency evaluation results at the 12 months (± 1 month) follow-up visit after the filling procedure

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Retention and fractures of the filling | ********************* | 3/3/3/ (3/3/3/) | 37 37373737 | 37 37373737 |
| Cases (Nmiss) A. No marginal fractures of the | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| filling | XXX (XX.X%) | XXX (XX.X%) | | |
| B. Minor marginal fractures of the filling without exposed | , , | , | | |
| dentin, clinically acceptable; C. Marginal fractures of the filling with exposed dentin, | XXX (XX.X%) | XXX (XX.X%) | | |
| clinically unacceptable | XXX (XX.X%) | XXX (XX.X%) | | |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |
| Marginal fractures of the filling | VAN (VAN) | 3/3/3/ (3/3/3/) | 37 37373737 | 37.373737 |
| Cases (Nmiss) A. No marginal fractures of the | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| filling | XXX (XX.X%) | XXX (XX.X%) | | |
| B. Minor marginal fractures of | 1221 (1211175) | 1221 (2211170) | | |
| the filling without exposed | | | | |
| dentin, clinically acceptable; | XXX (XX.X%) | XXX (XX.X%) | | |
| C. Marginal fractures of the | | | | |
| filling with exposed dentin, clinically unacceptable | XXX (XX.X%) | VVV (VV V0/.) | | |
| NA | XXX (XX.X%) | XXX (XX.X%)<br>XXX (XX.X%) | | |
| Contour and marginal adaptation | 7474 (7474.7470) | $\mathcal{M}\mathcal{M}(\mathcal{M}\mathcal{M},\mathcal{M}^{\prime},0)$ | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| A. Intact contour and continuous probing between the filling | ` , | , | | |
| and tooth | XXX (XX.X%) | XXX (XX.X%) | | |
| B. Pits on the surface of the | | | | |
| filling and discontinuous | | | | |
| probing between the filling and tooth without exposed | | | | |
| dentin; | XXX (XX.X%) | XXX (XX.X%) | | |
| C. Severe attrition and dents on | 1221 (1211175) | 1221 (2211170) | | |
| the surface of the filling with | | | | |
| exposed dentin, or probes | | | | |
| hooked at the margins of the | | ****** /**** *** ** | | |
| filling | XXX (XX.X%) | XXX (XX.X%) | | |
| NA | XXX (XX.X%) | XXX (XX.X%) | | |

Notes: 1. Likelihood  $\chi$ 2 test or Fisher's exact probability test will be used for group comparison of qualitative measures.

2. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 46 (FAS) Analysis results of X-ray examination results before and after the filling procedure

| Measures | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| X-ray (periapical radiograph) examination | n immediately after th | ne filling procedure | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal X-ray findings after the filling | | , | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| X-ray (periapical radiograph) examination | | | lure | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal or normal X-ray findings 1 wee | ek (± 3 days) after the | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| X-ray (periapical radiograph) examination | n 1 year ( $\pm$ 1 month) | after the filling proce | dure | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal X-ray findings 1 year (± 1 mor | nth) after the filling pr | rocedure | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| No | XXX (XX.X%) | XXX (XX.X%) | | |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| X-ray examination (screening→immediat | ely after the filling pr | rocedure) | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal→Abnormal | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal→Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal→Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal→Abnormal | XXX (XX.X%) | XXX (XX.X%) | | |
| X-ray examination (screening→1 week as | fter the filling proced | ure) | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal→Abnormal | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal→Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal→Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal→Abnormal | XXX (XX.X%) | XXX (XX.X%) | | |
| X-ray examination (screening→1 year aft | er the filling procedu | re) | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Normal→Abnormal | XXX (XX.X%) | XXX (XX.X%) | | |
| Normal→Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal→Normal | XXX (XX.X%) | XXX (XX.X%) | | |
| Abnormal→Abnormal | XXX (XX.X%) | XXX (XX.X%) | | |

<sup>2.</sup> Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

## Table 47 (FAS) Detailed descriptions of device defects

| Center code | Randomization No. | Group | | U | Applicable items at to a device defect | device defect | No. | Name of device defect | | | device defect | | Measures<br>taken | Any resulting medical events, diseases or injuries | 1 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XX | XXX | XX | XX | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XX | XXX | XX | XX | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XX | XXX | XX | XX | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Notes: 1. Treatment group:  $3M^{TM}$  Filtek $^{TM}$  Bulk Fill Posterior Restorative; Control group:  $3M^{TM}$  Filtek $^{TM}$  Z350XT.

Table 48 (FAS) (AE) Case specific descriptions of adverse event

| Center code | Randomization<br>No. | Group | Sex | Age | Name<br>of AE | Occurrence<br>time after the<br>procedure<br>(days) | Remission<br>time (days) | Characteristics of AE | Number of paroxysmal attacks | Severity | and report | Relationship to the investigational device | Outcomes | Sequela | Corrective treatment | Withdrawal from the trial | Serious<br>Adverse<br>Event |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XX | XXX | XX | XX | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XX | XXX | XX | XX | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XX | XXX | XX | XX | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Notes: 1. Occurrence time after the procedure = starting date of AE - date of cavity filling; Remission time = ending date of AE - starting date of AE; 2. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 49 (FAS) (AE) Summary of adverse events

| AEs | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Total number of AEs XXXX | XXX<br>XXX | XXX<br>XXX | | |
| Total cases of AEs Cases (Nmiss) Yes No | XXX (XXX)<br>XXX (XX.X%)<br>XXX (XX.X%) | XXX (XXX)<br>XXX (XX.X%)<br>XXX (XX.X%) | X.XXXX | X.XXXX |

- Notes: 1. The total cases of AEs refer to the number of subjects with AEs. A subject with one occurrence of AE will be deemed as "Yes".
  - 2. Likelihood  $\chi 2$  test or Fisher's exact probability test will be used for group comparison of qualitative measures.
  - 3. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 50 (FAS) Case specific descriptions of adverse events related to the investigational device

| Center code | Randomization<br>No. | Group | Sex | Age | Name<br>of AE | Occurrence<br>time after the<br>procedure<br>(days) | Remission<br>time (days) | Characteristics of AE | Number of paroxysmal attacks | Severity | and report | Relationship to the investigational device | Outcomes | Sequela | Corrective treatment | Withdrawal from the trial | Serious<br>Adverse<br>Event |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XX | XXX | XX | XX | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XX | XXX | XX | XX | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XX | XXX | XX | XX | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Notes: 1. AEs related to the investigational device refer to AEs that are "possibly related" or "quite possibly related" or "definitely related" to the investigational device.

<sup>2.</sup> Occurrence time after the procedure = starting date of AE - date of cavity filling; Remission time = ending date of AE - starting date of AE; 3. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 51 (FAS) Summary of adverse events related to the investigational device

| AEs | Treatment group | Control group | Statistics | P value |
|---------------------|-----------------|---------------|------------|---------|
| Total number of AEs | XXX | XXX | | |
| XXXX | XXX | XXX | | |
| ······ | | | | |
| Total cases of AEs | | | | |
| Cases (Nmiss) | XXX (XXX) | XXX (XXX) | X.XXXX | X.XXXX |
| Yes | XXX (XX.X%) | XXX (XX.X%) | | |
| No | XXX (XX.X%) | XXX (XX.X%) | | |

- Notes: 1. The total cases of AEs refer to the number of subjects with AEs. A subject with one occurrence of AE will be deemed as "Yes".
  - 2. Likelihood  $\chi 2$  test or Fisher's exact probability test will be used for group comparison of qualitative measures.
  - 3. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 52 (FAS) (SAE) Case specific descriptions of serious adverse events

| Center F | Randomizatio<br>No. | | Sex | Age | Name<br>of SAE | Occurrence<br>time after the<br>procedure<br>(days) | Remission<br>time (days) | Characteristic | Number of cs paroxysmal attacks | Severity | Relationship<br>to the<br>investigational<br>device | | Sequela | | Withdrawal from the trial | | | Report situations |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XX<br>XX | XXX<br>XXX | XX<br>XX | XX<br>XX | XX<br>XX | XXX<br>XXX | XXX<br>XXX | XXX<br>XXX | XXX | XXX<br>XXX | XXX<br>XXX | XXX<br>XXX | XXX<br>XXX | XXX<br>XXX | XXX | XXX<br>XXX | XXX<br>XXX | XXX | XXX |
| XX | XXX | XX | XX | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Notes: 1. Occurrence time after the procedure = starting date of SAE - date of cavity filling; Remission time = ending date of SAE - starting date of SAE; 2. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 53 (FAS) (SAE) Summary of serious adverse events

| Serious Adverse Event | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Total number of SAEs XXXX | XXX<br>XXX | XXX<br>XXX | | |
| Total cases of SAEs Cases (Nmiss) Yes No | XXX (XXX)<br>XXX (XX.X%)<br>XXX (XX.X%) | XXX (XXX)<br>XXX (XX.X%)<br>XXX (XX.X%) | X.XXXX | X.XXXX |

- Notes: 1. The total cases of SAEs refer to the number of subjects with SAEs. A subject with one occurrence of SAE will be deemed as "Yes".
  - 2. Likelihood  $\chi 2$  test or Fisher's exact probability test will be used for group comparison of qualitative measures.
  - 3. Treatment group:  $3M^{TM}$  Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 54 (FAS) Case specific descriptions of serious adverse events related to the investigational device

| Center l | Randomization<br>No. | | Sex | Age | Name<br>of SAE | Occurrence<br>time after the<br>procedure<br>(days) | | Characteristics<br>of SAE | Number of paroxysmal attacks | Severity | Relationship<br>to the<br>investigational<br>device | | Sequela | | Withdrawal from the trial | | | Report situations |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XX | XXX | XX | XX | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XX | XXX | XX | XX | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XX | XXX | XX | XX | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| •••• | | | | | | | | | | | | | | | | | | |

Notes: 1. SAEs related to the investigational device refer to SAEs that are "possibly related" or "quite possibly related" or "definitely related" to the investigational device.

<sup>2.</sup> Occurrence time after the procedure = starting date of SAE - date of cavity filling; Remission time = ending date of SAE - starting date of SAE; 3. Treatment group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 55 (FAS) Summary of serious adverse events related to the investigational device

| Serious Adverse Event | Treatment group | Control group | Statistics | P value |
|---|---|---|---|---|
| Total number of SAEs XXXX | XXX<br>XXX | XXX<br>XXX | | |
| Total cases of SAEs Cases (Nmiss) Yes No | XXX (XXX)<br>XXX (XX.X%)<br>XXX (XX.X%) | XXX (XXX)<br>XXX (XX.X%)<br>XXX (XX.X%) | X.XXXX | X.XXXX |

- Notes: 1. The total cases of SAEs refer to the number of subjects with SAEs. A subject with one occurrence of SAE will be deemed as "Yes".
  - 2. Likelihood  $\chi 2$  test or Fisher's exact probability test will be used for group comparison of qualitative measures.
  - 3. Treatment group:  $3M^{TM}$  Filtek<sup>TM</sup> Bulk Fill Posterior Restorative; Control group: 3M<sup>TM</sup> Filtek<sup>TM</sup> Z350XT.

Table 56 (FAS) List of subjects using concomitant drugs

| Center code | Randomization<br>No. | n<br>Group | Sex | Age | Drug name | Starting date | Ending time | Still in use | Administration route | n<br>Dosage | Unit | Indications | Justifications for treatment |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XX | XXX | XX | XX | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XX | XXX | XX | XX | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XX | XXX | XX | XX | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |